

Title: multicenter, randomized, double-blinded, placebo-controlled, parallel-group study to evaluate the efficacy, safety, and pharmacokinetics of intravenous MLN0002 (300 mg) infusion in induction and maintenance therapy in Japanese subjects with moderate or severe Crohn's disease

NCT Number: NCT02038920

Protocol Approve Date: 11-Nov-2013

Certain information within this protocol has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

# TAKEDA PHARMACEUTICALS PROTOCOL

## <Title>

Phase 3, multicenter, randomized, double-blinded, placebo-controlled, parallel-group study to evaluate the efficacy, safety, and pharmacokinetics of intravenous MLN0002 (300 mg) infusion in induction and maintenance therapy in Japanese subjects with moderate or severe Crohn's disease

## <Short Title>

# Phase 3 study of MLN0002 (300 mg) in treatment of Crohn's disease

**Sponsor:** Takeda Pharmaceutical Company Limited

1-1, Doshomachi 4-chome, Chuo-ku, Osaka-shi, Osaka

Study Number: MLN0002/CCT-001

**Version Number:** Initial version

IND Number: Not Applicable EudraCT Number: Not Applicable

Compound: Vedolizumab

Date: November 11, 2013

## CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered. Furthermore, the information is only meant for review and compliance by the recipient, his or her staff, and applicable institutional review committee and regulatory agencies to enable conduct of the study.

# 1.0 ADMINISTRATIVE INFORMATION AND PRINCIPLES OF CLINICAL STUDIES

1.1 Contacts and Responsibilities of Study-Related Activities

See the Annex.

# 1.2 Principles of Clinical Studies

This study will be conducted with the highest respect for the individual participants in accordance with the requirements of this study protocol and also in accordance with the following:

- The ethical principles that have their origin in the Declaration of Helsinki.
- International Conference on Harmonisation E6 Good Clinical Practice: Consolidated Guideline.
- All applicable laws and regulations, including, without limitation, data privacy laws, clinical trial disclosure laws, and regulations.

# **TABLE OF CONTENTS**

| 1.0 | | INISTRATIVE INFORMATION AND PRINCIPLES OF CLINICAL | |
|-----|-------|-----------------------------------------------------------|----|
| 1. | | ontacts and Responsibilities of Study-Related Activities | |
| 1 | | rinciples of Clinical Studies | |
| 2.0 | | DY SUMMARY | |
| 3.0 | | OF ABBREVIATIONS | |
| 3. | | efinitions in the Study | |
| 4.0 | | ODUCTION | |
| 4. | 1 Ba | ackground | 17 |
| 4. | 2 O | utcome of Clinical Studies | 17 |
| | 4.2.1 | Summary of Outcome of Phase 1 and 2 Studies Outside Japan | 18 |
| | 4.2.2 | Summary of Outcome of Phase 3 Studies Outside Japan | |
| | 4.2.3 | Summary of Outcome of Phase 1 Study in Japan | 19 |
| 4. | 3 Ra | ationale for the Proposed Study | 19 |
| 5.0 | STUL | OY OBJECTIVES AND ENDPOINTS | 20 |
| 5. | 1 O | bjectives | 20 |
| | 5.1.1 | Primary Objective for the Induction Phase | 20 |
| | 5.1.2 | Secondary Objective for the Induction Phase | 20 |
| | 5.1.3 | Primary Objective for the Maintenance Phase | 20 |
| | 5.1.4 | Secondary Objective for the Maintenance Phase | 20 |
| 5. | 2 E1 | ndpoints | 20 |
| | 5.2.1 | Efficacy Endpoints for the Induction Phase | 20 |
| | 5. | 2.1.1 Primary Endpoint | 20 |
| | 5. | 2.1.2 Secondary Endpoints | 20 |
| | 5. | 2.1.3 Exploratory Endpoints | 20 |
| | 5.2.2 | Efficacy Endpoints for the Maintenance Phase | 21 |
| | 5. | 2.2.1 Primary Endpoint | 21 |
| | 5. | 2.2.2 Secondary Endpoints | 21 |
| | 5. | 2.2.3 Exploratory Endpoints | 21 |
| | 5.2.3 | Pharmacokinetic Endpoint | 21 |
| | 5.2.4 | Safety Endpoints | 21 |
| | 5.2.5 | Immunogenicity Endpoint | 22 |
| 6.0 | STUE | DY DESIGN AND DESCRIPTION | 23 |
| 6. | 1 St | tudy Design | 23 |

| | 6.2 | | Jus | tification for Study Design, Dose, and Endpoints | 25 |
|---|---|---|---|---|---|
| | | 6.2 | .1 | Justification for Study Population | 25 |
| | | 6.2 | .2 | Justification of Study Design and Sample Size | 26 |
| | | 6.2 | .3 | Justification of the Placebo Group | 26 |
| | | 6.2 | .4 | Justification of the Dosage and the Evaluation Period | 26 |
| | | 6.2 | .5 | Justification of Endpoints | |
| | 6.3 | | Pre | mature Termination or Suspension of Study or Investigational site | 27 |
| | | 6.3 | .1 | Criteria for Premature Termination or Suspension of the Study | 27 |
| | | 6.3 | .2 | Criteria for Premature Termination or Suspension of Investigational Sites | 28 |
| | | 6.3 | .3 | Procedures for Premature Termination or Suspension of the Study or the Participation of Investigational Site(s) | 28 |
| 7.0 | ) | SEI | LEC | CTION AND DISCONTINUATION/WITHDRAWAL OF SUBJECTS | 29 |
| | 7.1 | | Inc | lusion Criteria | 29 |
| | 7.2 | | Exc | clusion Criteria | 30 |
| | 7.3 | | Exc | cluded Medications and Treatments | 33 |
| | | 7.3 | .1 | Rescue Treatments | 35 |
| | | 7.3 | .2 | Dose Reduction Schedule of Corticosteroids | 35 |
| | 7.4 | | Sul | oject Management | 36 |
| | 7.5 | | Cri | teria for Discontinuation or Withdrawal of a Subject | 37 |
| | 7.6 | | | cedures for Discontinuation or Withdrawal of a Subject | |
| 8.0 | ) | CL | INI | CAL STUDY MATERIAL MANAGEMENT | 39 |
| | 8.1 | | Stu | dy Medication and Materials | 39 |
| | | 8.1 | .1 | Dosage Form, Manufacturing, Packaging, and Labeling | 39 |
| | | | 8.1 | .1.1 Study Drug | 39 |
| | | | 8.1 | .1.2 Materials | 40 |
| | | 8.1 | .2 | Storage | 41 |
| | | 8.1 | .3 | Dose and Regimen | 41 |
| | | 8.1 | .4 | Overdose | 41 |
| | 8.2 | | Pro | cedures for Allocation, Prescription and Infusion of Study Drugs | 42 |
| | 8.3 | | | paration and Retention of the Allocation Table | |
| | 8.4 | | | servation of Blindness | |
| | 8.5 | | Pro | cedures for Blind-Breaking | 42 |
| | 8.6 | | Co | ntrol and Disposal of Sponsor-Supplied Drugs | 43 |
| 9.0 | ) | ST | | Y PLAN | |
| | 9.1 | | Stu | dy Procedures | 44 |

| | 9.1.1 | Informed Consent Procedure | 44 |
|---|---|---|---|
| | 9.1.2 | Demographics, Medical History, and Medication History Procedure | 44 |
| | 9.1.3 | Physical Examination Procedure | 45 |
| | 9.1.4 | Weight, Height and BMI | 45 |
| | 9.1.5 | Vital Sign Procedure | |
| | 9.1.6 | Documentation of Concomitant Medications and Non-drug Therapy | 46 |
| | 9.1.7 | Documentation of Concurrent Medical Conditions | 46 |
| | 9.1.8 | The Patient Diary | 46 |
| | 9.1.9 | CDAI Score | 47 |
| | 9.1 | .9.1 Calculation of Hematocrit (Ht) level scores | 48 |
| | 9.1.10 | Inflammatory Bowel Disease Questionnaire (IBDQ) | 48 |
| | 9.1.11 | Laboratory Test | 48 |
| | 9.1.12 | Contraception and Pregnancy Avoidance Procedure | 50 |
| | 9.1.13 | Pregnancy | 50 |
| | 9.1.14 | ECG Procedure | 51 |
| | 9.1.15 | PML Evaluation. | 51 |
| | 9.1.16 | Tuberculosis test | 51 |
| | 9.1.17 | Chest Imaging Procedure | 51 |
| | 9.1.18 | Pharmacogenomic Sample Collection | 51 |
| | 9.1.19 | Pharmacokinetic Sample Collection and Analysis | 52 |
| | 9.1.20 | Sample Collection for the HAHA/Neutralizing Antibody Test | 52 |
| | 9.1.21 | Record of Subjects Who Withdrew during the Screening Phase | 52 |
| | 9.1.22 | Enrollment into the induction Phase | 53 |
| | 9.1.23 | Registration of the Results of the Primary Efficacy Endpoint in the Induction Phase/Enrollment into the Maintenance Phase | 53 |
| | 9.1.24 | Enrollment into the Open-label Cohort | 53 |
| 9.2 | Stu | udy Drug Compliance | 54 |
| 9.3 | Sc | hedule of Observations and Procedures | 54 |
| | 9.3.1 | The Screening Phase (Visit 1) | 54 |
| | 9.3.2 | Induction Phase | 55 |
| | 9.3 | 3.2.1 Baseline Evaluation/Enrollment into the induction Phase (Visit 2) | 55 |
| | 9.3 | 3.2.2 Administration in the Induction Phase (Visits 3 and 4) | 56 |
| | 9.3 | 8.2.3 Evaluation of Primary Efficacy Endpoint (Visit 5)/Withdrawal during the | |
| | | Induction Phase | |
| | 9.3.3 | Maintenance Phase | 57 |

| 9.3.3.1 Enrollment into the maintenance Phase (Visit 6) | 57 |
|---|---|
| 9.3.3.2 Administration in the Maintenance Phase (Visits 7 through 1 | 7)57 |
| 9.3.3.3 Evaluation of Primary Efficacy Endpoint in the Maintenance (Visit 18)/Withdrawal during the Maintenance Phase | |
| 9.3.4 Open-label Cohort | 58 |
| 9.3.4.1 Enrollment into the open-label cohort (Visit 1x) | 58 |
| 9.3.4.2 Administration in the Open-label Cohort (Visits 2x through 2 | 24x)59 |
| 9.3.4.3 The Final Evaluation of the Open-label Cohort (VIST 25x)/V during the Open-label Cohort | |
| 9.3.5 The Unscheduled Visits | |
| 9.3.6 Predefined Study Completion | 60 |
| 9.3.7 At 16 weeks after the Last Dose | |
| 9.3.8 Post Study Care | 61 |
| 9.4 Retention and Disposal of Biological Samples | 61 |
| 9.5 Follow-Up Survey | 61 |
| 10.0 PRETREATMENT EVENTS AND ADVERSE EVENTS | 63 |
| 10.1 Definitions | 63 |
| 10.1.1 PTEs | 63 |
| 10.1.2 AEs | 63 |
| 10.1.3 Additional Points to Consider for PTEs and AEs | 63 |
| 10.1.4 SAEs | 65 |
| 10.1.5 Intensity of PTEs and AEs | 66 |
| 10.1.6 Causality of AEs | 66 |
| 10.1.7 Relationship to Study Procedures | |
| 10.1.8 Start Dates | 67 |
| 10.1.9 Stop Date | 67 |
| 10.1.10 Frequency | |
| 10.1.11 Action Concerning Study Drug | |
| 10.1.12 Outcome | |
| 10.2 Procedures | |
| 10.2.1 Collection and Reporting of AEs | |
| 10.2.1.1 PTE and AE Collection Period | |
| 10.2.1.2 PTE and AE Reporting | |
| 10.2.2 Collection and Reporting of SAEs | 69 |

| | 10.2.3 Drug-induced Liver Function Test Abnormal Possibly Leading to Sever Liver Disorder | |
|---|---|---|
| 10 | | |
| 10 | 10.3.1 SAE Reports to Investigators, the IRBs and Regulatory Authorities | |
| 11.0 | STUDY-SPECIFIC COMMITTEES | |
| _ | | |
| 11 | | |
| 12.0 | DATA HANDLING AND RECORDKEEPING | |
| 12 | 1 / | |
| 12 | | |
| 13.0 | | |
| 13 | J | |
| | 13.1.1 Analysis Sets | |
| | 13.1.2 Analysis of Demographics and Other Baseline Characteristics | |
| | 13.1.3 Efficacy Analysis | |
| | 13.1.4 Pharmacokinetic Analysis | |
| | 13.1.5 Safety Analysis | |
| | 13.1.6 Analysis of Immunogenicity Endpoints | |
| 13 | j , | |
| 13 | .3 Determination of Sample Size | 80 |
| 14.0 | QUALITY CONTROL AND QUALITY ASSURANCE | 81 |
| 14 | .1 Study-Site Monitoring Visits | 81 |
| 14 | .2 Protocol Deviations | 81 |
| 14 | .3 Quality Assurance Audits and Regulatory Agency Inspections | 81 |
| 15.0 | ETHICAL ASPECTS OF THE STUDY | 82 |
| 15 | .1 IRB Approval | 82 |
| 15 | | |
| 15 | | |
| 15 | .4 Publication, Disclosure, and Clinical Trial Registration Policy | 84 |
| | 15.4.1 Publication and Disclosure | |
| | 15.4.2 Clinical Trial Registration | |
| | 15.4.3 Clinical Trial Results Disclosure | |
| 15 | | |
| 16.0 | REFERENCES | |

| LIST OF IN- | TEXT TABLES | |
|---|---|---|
| Table 7.a | List of Excluded Drugs and Treatments | 33 |
| Table 8.a | Study drug | 39 |
| Table 8.b | Materials | 40 |
| Table 8.c | Dose and Regimen | 41 |
| Table 9.a | CDAI Scoring System for the Assessment of CD Activity [13] | 47 |
| Table 9.b | Laboratory tests | |
| Table 10.a | Takeda Medically Significant AE List | 66 |
| LIST OF IN- | TEXT FIGURES | |
| Figure 6.a | Schematic of Study Design | 24 |
| Figure 6.b | Schematic of Enrollments, Administrations, and Visits | 25 |
| Figure 8.a | Labels on Vials | 39 |
| Figure 8.b | A Label on Outer Packages | 40 |
| LIST OF AP | PENDICES | |
| Appendix A | Schedule of Study Procedures | 88 |
| Appendix B | Responsibilities of the Investigator | 92 |
| Appendix C | Diagnostic Criteria for CD (Revised on January 17, 2013) | 93 |
| Appendix D | PML Checklists | 98 |
| Appendix E | Follow-Up Survey Form | 103 |

## 2.0 STUDY SUMMARY

| Sponsor: | Compound: | |
|---|---|---|
| Takeda Pharmaceutical Company Limited | MLN0002 | |
| Study title: Phase 3, multicenter, randomized, double-blinded, | IND No.: | EudraCT No.: |
| placebo-controlled, parallel-group study to evaluate the | Not Applicable | Not Applicable |
| efficacy, safety, and pharmacokinetics of intravenous | | |
| MLN0002 (300 mg) infusion in induction and maintenance | | |
| therapy in Japanese subjects with moderate or severe Crohn's | | |
| disease | | |
| Study Number: MLN0002/CCT-001 | Phase :3 | |

### **Study Design:**

This is a phase 3, multicenter, randomized, double-blinded, placebo-controlled, parallel-group study to evaluate the efficacy, safety, and pharmacokinetics of MLN0002 in induction and maintenance therapies in Japanese subjects with moderate or severe Crohn's disease (CD). This study consists of the screening, induction and maintenance phases, and the open-label cohort.

The screening phase involves screening tests of consenting subjects who visit a study site between 21 and 7 days before the start of treatment. Subjects meeting the eligibility criteria based on the inclusion and exclusion criteria on the first day of treatment (Day 1) will be enrolled into the induction phase.

Subjects enrolled into induction phase will be randomized 1:1 to the placebo or MLN0002 group to receive the placebo or 300 mg of MLN0002 at Weeks 0, 2, and 6 in a double-blinded manner. The primary efficacy endpoint in the induction phase will be evaluated at Week 10.

Subjects showing a CDAI-70 response to the study drug at Week 10 will be enrolled into the maintenance phase at Week 14. Subjects who received the placebo in the induction phase will continue to receive the placebo at Weeks 14, 22, 30, 38, 46, and 54 in a double-blinded manner. Subjects who received MLN0002 in the induction phase will be randomized 1:1 to the placebo or MLN0002 group, and will receive the placebo or 300 mg of MLN0002 at Weeks 14, 22, 30, 38, 46, and 54 in a double-blinded manner. The primary efficacy endpoint in the maintenance phase will be evaluated at Week 60.

Subjects not showing a CDAI-70 response to the study drug at Week 10 can be enrolled into the open-label cohort. Setting the enrollment day to the open-label cohort as Week 0x, those subjects will receive 300 mg of MLN0002 at Weeks 0x, 2x, 6x and then every 8 weeks thereafter for 46 weeks (minimum) to 94 weeks (maximum) in an unblinded manner. Subjects who experienced disease worsening or received rescue treatments during the maintenance phase, or those who completed Week 60 of the maintenance phase can be enrolled into the open-label cohort to receive the study drug in the same manner. Administration of MLN0002 will be terminated in all subjects at Week 46x of the last subject enrolled into the open-label cohort.

The end-of-study examination will be performed at 16 weeks after the last dose in all subjects who received the study drug. In addition, the follow-up survey will be performed every 6 months from the last dose of the study drug up to 2 years or until the date of marketing approval of the study drug, whichever comes earlier.

### Primary objective for the induction phase:

To evaluate efficacy of MLN0002 in induction therapy in Japanese subjects with moderate or severe CD.

## Secondary objective for the induction phase:

To evaluate safety of MLN0002 in induction therapy in Japanese subjects with moderate or severe CD.

## Primary objective for the maintenance phase:

To evaluate efficacy of MLN0002 in maintenance therapy in Japanese subjects with moderate or severe CD.

### **Secondary objective for the maintenance phase:**

To evaluate safety of MLN0002 in maintenance therapy in Japanese subjects with moderate or severe CD.

| Subjects: Japanese subjects with moderate or severe CD | |
|---|---|
| Number of Subjects: | Number of Sites: |
| Approximately 110 in total. | Approximately 60 sites |
| Maximum 152 subjects. The target number of | |
| subjects without a history of anti-TNFα antibody | |
| therapy is approximately 25% of the total. | |
| Dose Level(s): | Route of Administration: |
| MLN0002 (300 mg) or the placebo will be | Intravenous infusion (IV) |
| administered by intravenous infusion at Weeks 0, | |
| 2, 6 and every 8 weeks thereafter. | |
| Duration of Treatment: | Period of Evaluation: |
| 54 weeks (maximum 154 weeks) | 70 weeks (maximum 170 weeks) |
| | The follow-up survey will be performed every 6 months from the |
| | last dose of the study drug for up to 2 years or until the date of |
| | marketing approval of the study drug, whichever comes earlier. |

#### **Main Criteria for Inclusion:**

- Subjects aged 15 to 80 (inclusive) at the time of signing the informed consent.
- Subjects with any diagnosis of the small intestine type, the large intestine type or the small/large intestine type of CD based on the Revised Diagnostic Criteria for CD issued by Research Group for Intractable Inflammatory Bowel Disease Designated as Specified Disease by the Ministry of Health, Labor and Welfare (MHLW) of Japan (2012) at least 3 months before start of administration of the study drug.
- Subjects with a CDAI score of 220≤ and ≤450 points at the first dose of the study drug, and also meeting any of the following:
  - Subjects with a CRP level of >0.30 mg/dL at the screening test.
  - Subjects confirmed to have irregular-to-round shaped ulcers or multiple aphtha in the small or large intestine extensively (≥10 lesions) in the endoscopy or the imaging test within 4 month before the first dose of the study drug.
  - Subjects confirmed to have longitudinal ulcers or a cobblestone appearance in the small or large intestine in the endoscopy or the imaging test within 4 months before the first dose of the study drug.
- Subjects whose complication of colon cancer or dysplasia had to be ruled out by total colonoscopy at the start of the study drug administration (or the results from total colonoscopy performed within 1 year before giving consent are available), if subjects met any of the followings; subjects with extensive or limited colitis of ≥8 years duration, subjects aged ≥50 years, or subjects with a first-degree family history of colon cancer.
- Subjects meeting the following treatment failure criteria with at least one of the following agents within 5 year before signing the informed consent:

Corticosteroids

- Resistance
- Dependence
- Intolerance

Immunomodulators [azathioprine (AZA), 6-mercaptopurine (6-MP) or methotrexate (MTX)]

- Refractory
- Intolerance

Anti-TNFα antibodies

- Inadequate response
- Loss of response
- Intolerance

#### Main Criteria for Exclusion:

- Subjects who have or are suspected of having abdominal abscess.
- Subjects with a history of subtotal or total colectomy.
- Subjects with a history of  $\geq 3$  enterectomy, or a history of diagnosis of short bowel syndrome.
- Subjects with ileostomy, colostomy, or internal fistula or severe intestinal stenosis.
- Subjects who started an oral 5-aminosalicylic acid (5-ASA), probiotics treatment, an antibiotic for CD treatment, or an oral corticosteroid of ≤30 mg/day within 13 days before the first dose of the study drug. Subjects who have used these drugs for at least 14 days before the first dose of the study drug, and who changed dosage of or discontinued these drugs within 13 days before the first dose of the study drug.
- Subjects who have received 5-ASAs, corticosteroid enemas/suppositories, corticosteroid IV infusion, oral corticosteroid at >30 mg/day, drugs for diarrhea-predominant irritable bowel syndrome, or Chinese herbal medicine for the treatment of CD (e.g., Daikenchuto) within 13 days before the first dose of the study drug.
- Subjects who have used AZA, 6-MP or MTX within 27 days before the first dose of the study drug However, this will not apply to subjects who have used these drugs for 83 or more days before the first dose of the study drug and continued the steady dose administration of the drugs for 27 or more days before the first dose of the study drug.
- Subjects who have received cyclosporine, tacrolimus, tofacitinib or any study drugs of low-molecular compound for CD treatment within 27 days before the first dose of the study drug.
- Subjects who have received adalimumab within 27 days before the first dose of the study drug or any biological drugs other than adalimumab within 55 days before the first dose of the study drug However, this will not apply to subjects who have topically received these drugs (e.g., intraocular injection for treatment of age-related macular degeneration).
- Subjects who have received any live-vaccinations within 27 days before the first dose of the study drug
- Subjects who underwent an enterectomy within 27 days before the first dose of the study drug or those anticipated to require an enterectomy during the study.
- Subjects who have received leukocytapheresis or granulocyte apheresis within 27 days before the first dose of the study drug.
- Subjects who received central venous nutrition therapy or enteral total nutrition therapy, or fasted within 20 days before the first dose of the study drug.
- Subjects who received an enteral nutrient of >900 kcal/day or who will begin to receive an enteral nutrient of ≤900 kcal/day within 20 days before the first dose of the study drug. Subjects who had received an enteral nutrient of ≤900 kcal/day earlier than 21 days before the first dose of the study drug, and modified or discontinued the dosage within 20 days before the first dose of the study drug.
- Subjects with an evidence of adenomatous colonic polyps that need to be removed at the start of study drug administration.
- Subjects with a history or a complication of large or small intestinal dysplasia.

## Main efficacy endpoints of the induction phase:

## Primary endpoint:

CDAI-100 response at Week 10

## Secondary endpoints:

Clinical remission at Week 10

Change in CRP level over time in the subpopulation of subjects with the baseline CRP level of >0.30 mg/dL

### Main efficacy endpoints of the maintenance phase:

## Primary endpoint:

Clinical remission at Week 60

#### Secondary endpoints:

CDAI-100 response at Week 60, durable remission in the maintenance phase, and corticosteroid-free remission at

Week 60

### Pharmacokinetic endpoints:

Serum MLN0002 concentration

## Safety endpoints:

Adverse events (AEs), body weight, vital signs, electrocardiogram (ECG), clinical laboratory test (blood biochemistry, hematology, and urinalysis)

### **Immunogenicity endpoints:**

HAHA, neutralizing antibody

# Statistical analysis plan:

(1) Statistical analysis in the induction phase

The following descriptive calculations will be performed in the "Full Analysis Set in the induction phase (subjects randomized and received the study drug at least once in the induction phase)."

For the primary efficacy analysis, "CDAI-100 response at Week 10" (primary endpoint of the induction phase) will be calculated by treatment group of the induction phase. Also CDAI-100 response at Week 10 will be calculated with stratification according to a history of anti-TNF $\alpha$  antibody therapy, and the comparison between treatment groups will be made with the Cochran-Mantel-Haenszel (CMH) test with 2-sided significance level of 10% by using a history of anti-TNF $\alpha$  antibody therapy as a stratification factor. The results of the primary analysis of the induction phase will be interpreted as below to determine the efficacy of MLN0002 induction therapy.

The superiority of MLN0002 over the placebo on CDAI-100 response at Week 10 in the primary analysis of the
induction phase is demonstrated when a statistically significant difference is observed in the CDAI-100 response
at Week 10.

For the secondary efficacy analysis, clinical remission at Week 10 will be calculated in the same manner as those in the primary analysis in the induction phase. The results of the secondary analysis will be interpreted as below to determine the efficacy of MLN0002 induction therapy.

- The superiority of MLN0002 over the placebo on clinical remission at Week 10 in the primary analysis of the induction phase is demonstrated when a statistically significant difference is observed in both the CDAI-100 response at Week 10 and clinical remission at Week 10.
- (2) Statistical analysis in the maintenance phase

The following descriptive calculations will be performed in the "Full Analysis Set of the maintenance phase (subjects randomized and received the study drug at least once in the maintenance phase)."

For the primary efficacy analysis, "clinical remission at Week 60" (primary endpoint of the maintenance phase)" will be calculated by treatment group of the maintenance phase.

### Sample size justification:

On the basis of findings from the phase 3 double-blinded, placebo-controlled study of MLN0002 induction therapy in non-Japanese moderate to severe CD subjects who had failed with an anti-TNF $\alpha$  antibody (C13011), the CDAI-100 response at Week 10 in MLN0002 and the placebo was estimated as 47.2% and 24.6%, respectively, clinical remission at Week 10 in MLN0002 and the placebo was estimated as 28.7% and 13.0%, respectively, and the CDAI-70 response at Week 10 in MLN0002 and the placebo was estimated as 56.9 % and 38.7%, respectively, in the study.

When the CDAI-100 response at Week 10 in the induction phase is analyzed using Pearson's chi-square test with 2-sided significance level of 10%, 55 subjects each (at a ratio of 1:1, total 110) will be required for the MLN0002 and placebo group to detect significance with a power of at least 80% for the MLN0002 and placebo group. Similarly, 76 subjects each (total 152) will be required to detect significance with a power of at least 90%. These numbers were therefore selected as the numbers of evaluable subjects of the primary endpoint of the induction phase (number of "subjects who were randomized in the induction phase and received at least one dose of the study drugs in the induction phase"). When the clinical remission at Week 10 is analyzed in the same manner on the accumulated 55 to 76 subjects to be evaluated for the primary endpoint in the induction phase, statistical significances in both the CDAI-100 response at Week 10 and clinical remission at Week 10 are detected with a power of 61 to 76%.

Number of subjects to be evaluated for the primary endpoint in the maintenance phase (number of subjects who were randomized and received at least one dose of the study drug in the maintenance phase) is 16 to 22 subjects in each group and 32 to 44 subjects in total based on the above estimation.

## 3.0 LIST OF ABBREVIATIONS

5-ASA 5-aminosalicylic acid 6-MP 6-mercaptopurine ALT alanine aminotransferase

ALP alkaline phosphatase
AST aspartate aminotransferase

AZA Azathioprine
BMI body mass index
BUN blood urea nitrogen
CD Crohn's disease

CDAI Crohn's Disease Activity Index

CRP C-reactive protein

ELISA Enzyme-Linked ImmunoSorbent Assay

FDA Food and Drug Administration

GCP Good Clinical Practice

γ-GTP γ-glutamyl transpeptidase

HAHA human anti-human antibody

HBs hepatitis B surface antigen

hCG human chorionic gonadotropine

HCV hepatitis C virus

HIV human immunodeficiency virus

Ht hematocrit

IBDQ Inflammatory Bowel Disease Questionnaire ICH International Conference on Harmonisation

INR International normalized ratio

MedDRA Medical Dictionary for Regulatory Activities

MHRA Medicines and Healthcare products Regulatory Agency

MTX methotrexate

PMDA Pharmaceutical and Medical Devices Agency
PML progressive multifocal leukoencephalopathy
SUSARs suspected serious unexpected adverse reactions

TNF Tumor Necrosis Factor

CD Ulcerative colitis

WHO World Health Organization

# 3.1 Definitions in the Study

The definitions in the study are provided below;

| Terms | Definitions |
|---|---|
| Clinical remission | CDAI score of ≤150 |
| CDAI-70 response | A ≥70-point decrease in CDAI score from baseline |
| CDAI-100 response | A ≥100-point decrease in CDAI score from baseline |
| Durable remission in the maintenance phase | Clinical remission at ≥80% of the scheduled visits including Week 60 |
| Durable CDAI-100 response in the maintenance phase | CDAI-100 response at ≥80% of the scheduled visits including Week 60 |
| Corticosteroid-free remission at Week 60 | Clinical remission with corticosteroid-free at Week 60, though corticosteroids were used at the first dose of the study drug |
| Disease worsening | In the maintenance phase, a $\geq$ 100-point increase in CDAI score from Week 10 value and CDAI score of $\geq$ 220 on 2 consecutive visits*, <b>OR</b> |
| | In the open-label cohort, a $\geq$ 100-point increase in CDAI score from Week 10x value and CDAI score of $\geq$ 220 on 2 consecutive visits* |
| Sustained non-response | CDAI-70 non-response during 20 weeks from the first dose of the study drug and CDAI score of ≥220 |
| Rescue medications | Any new medications, increases in dose of baseline medications, or new concomitant therapies required for treatment for unresolved CD symptom (except abscess drainage or the Seton method for the anal lesion) |
| | Note, however, that any increases in dose or beginning use of medications permitted in the open-label cohort, dosed after the subject was enrolled into the open-label cohort, were not regarded as the rescue medications |
| Treatment failure | Disease worsening, rescue medications, or withdrawal due to study drug-related AEs |

<sup>\*</sup> The 2 visits included the unscheduled visits due to CD worsening. The interval between visits was to be at least 1 week, where possible.

## 4.0 INTRODUCTION

# 4.1 Background

Crohn's Disease (CD) is a granulomatous inflammatory disease most commonly found in young people. The disease, affecting any part of the gastrointestinal tract from the mouth throughout the anus, forms characteristic conditions mainly in the small and large intestine such as intestinal stenosis and fistula with edema and ulcers. As various complications may be induced even outside the gastrointestinal tract, systemic symptoms including fever, weight loss or malnutrition, or complication-induced symptoms including anemia, arthritis, iritis or skin lesions may emerge in addition to gastrointestinal symptoms including diarrhea or abdominal pain. The disease condition may progress with repetition of recurrence and remission, and often become resistant to treatments to deteriorate social activity.

In the disease, it is believed that breakdown of the mucosal immune system by some genetic predisposition may lead to a exaggerated immune response against intraluminal antigens including enterobacteria or diet, resulting in progression and persistence of inflammation, however etiology is still unrevealed. A curative treatment has not been established, therefore treatment approaches aim to control disease activity with the remission induction therapy and the remission maintenance therapy in order to improve the Quality of Life (QOL). Possible treatment approaches including medical treatment (e.g., pharmacotherapy and nutrition therapy) and surgical treatment are detailed in line with the types and severities of the disease in the Revised Treatment Guideline (draft)[1] issued by "Research Group for Intractable Inflammatory Bowel Disease" Designated as Specified Disease by the MHLW of Japan.

MLN0002 is a recombinant human immunoglobulin  $G_1$  monoclonal antibody[2] that specifically binds to human lymphocyte  $\alpha_4\beta_7$  integrin, and is currently being developed in ulcerative colitis (UC) and CD inside/outside Japan.

MLN0002 binds and inhibits  $\alpha_4\beta_7$  integrin, a cell membrane protein of lymphocytes, to bind its principal ligand of mucosal addressin cell adhesion molecule-1 (MAdCAM-1; a transmembrane glycoprotein markedly expressing on vascular endothelial cells in the high endothelial venule in the Peyer patch or the mesenteric lymph node and the arteriole in the intestinal lamina propria), leading to suppression of lymphocytes to migrate toward the intestinal mucosa and the gut-related lymphoid tissue[2]. From the above, MLN0002 is anticipated to exert efficacy with superior safety to conventional treatments or other biological drugs in UC and CD through suppression of intestinal inflammation by gastrointestinal tract-selective immunomodulatory effect not requiring systemic immunosuppression[3][4].

## 4.2 Outcome of Clinical Studies

Outside Japan, the following 4 Phase 3 studies (GEMINI Programs) were conducted in subjects with UC and CD in addition to the 14 Phase 1 and 2 studies. As of October, 2013, all studies were completed except a long-duration study in subjects with UC and CD (C13008), and applications

have been submitted in Europe and US. In Japan, the Phase 1 study was conducted in subjects with UC.

| Study Number | Study Title |
|---|---|
| C13006 | Phase 3, double-blinded, placebo-controlled study of induction and maintenance therapies in moderate to severe UC patients (GEMINI 1). |
| C13007 | Phase 3, double-blinded, placebo-controlled study of induction and maintenance therapies in moderate to severe CD patients (GEMINI 2). |
| C13011 | Phase 3, double-blinded, placebo-controlled study of induction therapy in moderate to severe CD patients who had failed with anti-TNFα antibodies therapy (GEMINI 3). |
| C13008 | Phase 3, long-term open-label safety and efficacy study in UC or CD patients who had been enrolled in the Phase 2 and Phase 3 study of MLN0002. |

# 4.2.1 Summary of Outcome of Phase 1 and 2 Studies Outside Japan

Major outcomes in Phase 1 and 2 studies conducted outside Japan were summarized below;

- The pharmacokinetics of MLN0002 at the doses of 2 to 10 mg/kg was linear. The elimination half-life of MLN0002 was 15 to 22 days[5].
- The  $\alpha_4\beta_7$  receptors were saturated after the first dose at the doses of 2 to 10 mg/kg. Saturation of  $\alpha_4\beta_7$  receptors had been dose-dependently continued for several months after the last dose[5].
- It was suggested that the human anti-human antibody to MLN0002 (anti-MLN0002 antibody; hereinafter referred to as HAHA) may eliminate MLN0002 from the blood, resulting in decrease of MLN0002 exposure and loss of saturation of  $\alpha_4\beta_7$  receptors. HAHA emergence was dose-dependently decreased.
- MLN0002 demonstrated superiority to the placebo in all subjects as clinical remission was 32% at Week 6 in UC and 37% at Week 8 in CD[6][7]. The frequency of AEs was not significantly different from that in the placebo with no particular safety issues.

# 4.2.2 Summary of Outcome of Phase 3 Studies Outside Japan

In all 3 Phase 3 studies conducted outside Japan (C13006, C13007 and C13011), 300 mg of MLN0002 or the placebo were administered. In C13006 study, superiorities were demonstrated to the placebo in the primary endpoints, i.e., the clinical response in the induction phase and the clinical remission in the maintenance phase[8]. Two primary endpoints were set in the induction phase of C13007 study. The difference in the clinical response in CD Activity Index (CDAI)-100 was not significant, however superiority to the placebo was demonstrated in the clinical remissions each in the induction phase and the maintenance phase[9]. In C13011 study, superiority to the placebo was not demonstrated in the primary endpoint of the clinical remission at Week 6 in the sub-population of subjects who had failed with anti-TNFα antibodies (75% of all population), however the clinical remission at Week 6 in the whole population was significantly different from the placebo. In addition, the significant difference from the placebo in the clinical remission at

Week 10 was observed both in the sub-population who had failed an anti-TNF $\alpha$  antibody and the whole population[10].

Furthermore, incidence of AEs and serious adverse events (SAEs) were not significantly different between the whole MLN0002 group and placebo group. Progressive multifocal leukoencephalopathy (PML) was not observed in any subjects in completed or ongoing clinical development programs.

# 4.2.3 Summary of Outcome of Phase 1 Study in Japan

In Japan, the Phase 1 repeated-dose study in UC patients (CPH-001) was conducted to investigate safety, pharmacokinetics and pharmacodynamics of MLN0002 dosed at 150 or 300 mg in Weeks 0, 2 and 6. MLN0002 was well tolerated by the dose of 300 mg, and no injection site reaction or anaphylactic reaction was observed. In addition, serum MLN0002 concentration increased depending on dose ratio, and saturation of  $\alpha 4\beta 7$  receptors of the pharmacodynamic index was observed mostly continuously from the first dose[11].

# 4.3 Rationale for the Proposed Study

- In the 3 Phase 3 studies conducted outside Japan (C13006, C13007 and C13011), efficacy and safety of 300 mg of MLN0002 were investigated against the placebo each in the induction phase and the maintenance phase in moderate to severe UC or CD patients who had failed with the existing pharmacotherapy including anti-TNFα antibodies. As a result, significant difference from the placebo was observed in efficacy evaluation of MLN0002 in all studies. In addition, no particular issues were found in the safety evaluation. These results were consistent with the outcome obtained until Phase 2 studies.
- In Japan, safety, serum MLN0002 concentration and saturability of α4β7 receptors were investigated in UC patients dosed with 150 or 300 mg of MLN0002 at Weeks 0, 2 and 6. The serum MLN0002 concentration resulted in similarity inside/outside Japan, and saturation of α4β7 receptors was observed mostly continuously from the first dose. In addition, no safety issues were found.

From the above, the study was proposed as a Phase 3 study to investigate efficacy and safety of 300 mg of MLN0002 in moderate to severe Japanese CD patients.

Pharmacogenomic analysis may be conducted to evaluate contribution of genetic variance on drug response, for example, its efficacy and safety. Participation of study subjects in pharmacogenomic sample collection is optional.

As pharmacogenomics is an evolving science, currently many genes and their function are not yet fully understood. Future data may suggest a role of some of these genes in drug response or diseases, which may lead to additional hypothesis-generating exploratory research on banked samples.

## 5.0 STUDY OBJECTIVES AND ENDPOINTS

# 5.1 Objectives

# 5.1.1 Primary Objective for the Induction Phase

To evaluate efficacy of MLN0002 in induction therapy in Japanese subjects with moderate or severe CD.

# **5.1.2** Secondary Objective for the Induction Phase

To evaluate safety of MLN0002 in induction therapy in Japanese subjects with moderate or severe CD.

# 5.1.3 Primary Objective for the Maintenance Phase

To evaluate efficacy of MLN0002 in maintenance therapy in Japanese subjects with moderate or severe CD.

# 5.1.4 Secondary Objective for the Maintenance Phase

To evaluate safety of MLN0002 in maintenance therapy in Japanese subjects with moderate or severe CD.

# 5.2 Endpoints

## **5.2.1** Efficacy Endpoints for the Induction Phase

## 5.2.1.1 Primary Endpoint

• CDAI-100 response at Week 10

## 5.2.1.2 Secondary Endpoints

- Clinical remission at Week 10
- Change in CRP level over time in the subpopulation of subjects with the baseline CRP level of >0.30 mg/dL

# 5.2.1.3 Exploratory Endpoints

- Clinical remission at Week 6
- CDAI-100 response at Week 6
- CDAI-100 response at Week 6 and Week 10, and clinical remission at Week 6 and Week 10 in the sub-population of subjects without a history of anti-TNFα antibody therapy and in the sub-population of subjects who had failed with an anti-TNFα antibody therapy

- CDAI-100 response at Week 6 and Week 10, and clinical remission at Week 6 and Week 10 in the sub-population of subjects who had failed with a corticosteroid monotherapy and an immunomodulator (except those failed with an anti-TNFα antibody)
- IBDQ score change at Week 10 from baseline
- CDAI score change over time

# **5.2.2** Efficacy Endpoints for the Maintenance Phase

# 5.2.2.1 Primary Endpoint

• Clinical remission at Week 60

## 5.2.2.2 Secondary Endpoints

- CDAI-100 response at Week 60
- Durable remission in the maintenance phase
- Corticosteroid-free remission at Week 60

# 5.2.2.3 Exploratory Endpoints

- Clinical remission at Week 60 in the sub-population of subjects without a history of anti-TNFα antibody therapy and in the sub-population of subjects who had failed with an anti-TNFα antibody
- IBDQ score change at Week 38 and Week 60 from Week 14
- CDAI score change over time
- Change in CRP level over time in the subpopulation of subjects with the baseline CRP level of >0.30 mg/dL

# 5.2.3 Pharmacokinetic Endpoint

• Serum MLN0002 concentration

## 5.2.4 Safety Endpoints

- Adverse events (AEs)
- Body weight
- Vital signs
- ECG
- Clinical laboratory test (blood biochemistry, hematology and urinalysis)

## **CONFIDENTIAL**

# 5.2.5 Immunogenicity Endpoint

• HAHA, neutralizing antibody

# 6.0 STUDY DESIGN AND DESCRIPTION

# 6.1 Study Design

This is a phase 3, multicenter, randomized, double-blinded, placebo-controlled, parallel-group study to evaluate the efficacy, safety, and pharmacokinetics of MLN0002 in induction and maintenance therapies in Japanese subjects with moderate or severe CD. This study consists of the screening, induction, maintenance phases and open-label cohort.

The screening phase involves screening tests of consenting subjects who visit a study site between 21 and 7 days before the start of treatment. Subjects meeting the eligibility criteria based on the inclusion and exclusion criteria on the first day of treatment (Day 1) will be enrolled into the induction phase.

Subjects enrolled into induction phase will be randomized 1:1 to the placebo or MLN0002 group<sup>1</sup>, and will receive the placebo or 300 mg of MLN0002 at Weeks 0, 2, and 6 in a double-blinded manner. The primary efficacy evaluation in the induction phase will be performed at Week 10.

Subjects showing a CDAI-70 response to the study drug at Week 10 will be enrolled into the maintenance phase at Week 14. Subjects who received the placebo in the induction phase will continue to receive the placebo at Weeks 14, 22, 30, 38, 46, and 54 in a double-blinded manner. Subjects who received MLN0002 in the induction phase will be randomized 1:1 to the placebo or MLN0002 group<sup>2</sup> to receive the placebo or 300 mg of MLN0002 at Weeks 14, 22, 30, 38, 46 and 54 in a double-blinded manner. The primary efficacy endpoint in the maintenance phase will be evaluated at Week 60.

Subjects not showing a CDAI-70 response to the study drug at Week 10 can be enrolled into the open-label cohort. Setting the enrollment day to the open-label cohort as Week 0x, those subjects will receive 300 mg of MLN0002 at Weeks 0x, 2x, 6x and then every 8 weeks thereafter for 46 weeks (minimum) to 94 weeks (maximum) in an unblinded manner. Subjects who experienced disease worsening or received rescue treatments during the maintenance phase, or those who completed Week 60 of the maintenance phase can be enrolled into the open-label cohort to receive the study drug in the same manner. Administration of MLN0002 will be terminated in all subjects at Week 46x of the last subject enrolled into the open-label cohort.

The end-of-study examination will be performed at 16 weeks after the last dose in all subjects who received the study drug. In addition, the follow-up survey will be performed every 6 months from the last dose of the study drug up to 2 years or until the date of marketing approval of the study drug, whichever comes earlier (see Section 9.5).

Planned sample size is approximately 110 subjects in total and 152 subjects at maximum. In the situation, the number of subjects to be randomized in the induction phase is 55 to 76 in the

<sup>&</sup>lt;sup>1</sup>The dynamic allocation with the treatment history with anti-TNFα antibodies, concomitant use of an immunomodulator or corticosteroid, and the study sites.

 $<sup>^{2}</sup>$ The dynamic allocation with the treatment history with anti-TNFα antibodies, concomitant use of an immunomodulator or a corticosteroid, the study sites, and responder/non-responder at Week 10.

MLN0002 group and 55 to 76 in the placebo group. The target number of subjects without a history of anti-TNF $\alpha$  antibody therapy is approximately 25% of the total.

A schematic of the study design and a schematic of enrollments, administrations and visits are shown in Figure 6.a and Figure 6.b, respectively. A schedule of assessments is listed in Appendix A.

Figure 6.a Schematic of Study Design





Figure 6.b Schematic of Enrollments, Administrations, and Visits

W: Week, V: Visit

- a) CDAI-70 responders at Week 10 (evaluation of the primary efficacy endpoints in the induction phase) will be enrolled into the maintenance phase at Week 14. Non-CDAI-70 responders at Week 10 may be enrolled into the open-label cohort after completion of the Week 10 evaluation.
- b) Subjects who experienced disease worsening or received rescue treatments during the maintenance phase may be enrolled into the open-label cohort after completion of the evaluation at withdrawal of the maintenance phase. However, these subjects will be enrolled into the open-label cohort 3 to 9 weeks after the last dose in the maintenance phase.
- c) Subjects who completed Week 60 (evaluation of the primary efficacy endpoint in the maintenance phase) may be enrolled into the open-label cohort after completion of the Week 60 evaluation.

# 6.2 Justification for Study Design, Dose, and Endpoints

## **6.2.1** Justification for Study Population

The Guideline for Treatment of CD[1] issued by "Research Group for Intractable Inflammatory Bowel Disease Designated as Specified Disease" by the MHLW of Japan (2012) recommends 5-ASAs as the first line drug in the remission induction therapy in mild to moderate CD patients, and also recommends combination with the nutrition therapy in acceptable patients. Also, in moderate to severe patients, oral corticosteroids, antibiotics and immunomodulators are recommended in addition to the above treatments. Furthermore, anti-TNF $\alpha$  antibodies are recommended to non-responders to the remission induction therapy with corticosteroids or the nutrition therapy. However, poor response to anti-TNF $\alpha$  antibodies or loss of response during treatment with anti-TNF $\alpha$  antibodies are still problematic. MLN0002, having a different mode of action from existing therapeutic drugs, has been suggested to be efficacious in such patients by outcome from studies outside Japan.

From the above, the population in the induction phase in the study was set as moderate to severe Japanese CD patients who had failed with existing pharmacotherapy (any of corticosteroids/immunomodulators/anti-TNFα antibodies).

# 6.2.2 Justification of Study Design and Sample Size

The Guideline for Treatment of CD[1] recommends that the remission maintenance therapy should apply to prevent recurrence after achievement of remission induction. However, effective drugs in the induction therapy are not always efficacious in the maintenance therapy. The randomized, double-blinded, placebo-controlled study with an induction phase and maintenance phase was designed to objectively evaluate efficacy and safety both in the induction therapy and maintenance therapy. Additionally, the enrichment design was employed to evaluate efficacy and safety in the maintenance phase, in which only responders to MLN0002 in the induction phase will be enrolled in the population to be randomized in the maintenance phase.

For preservation of blindness, all responders at Week 10 will be enrolled into the maintenance phase irrespective of the drugs allocated in the induction phase. The responders who received MLN0002 in the induction phase will be randomized either to the placebo group or the MLN0002 group for evaluation of efficacy and safety of the maintenance therapy, and the responders who received the placebo in the induction phase will be continued to be allocated to the placebo groups.

In the ethically-established open-label cohort, it was designed that non-responders in the induction phase, patients who experienced disease worsening or received rescue treatments during the maintenance phase, or those completed Week 60 of the maintenance phase may continue to receive MLN0002 for 46 weeks (minimum) to 94 weeks (maximum).

See Section 13.3 for justification of the sample size.

## **6.2.3** Justification of the Placebo Group

Any active comparator is impossible to be used properly in the study in moderate to severe CD patients who had failed with existing pharmacotherapy (either of corticosteroids/immunomodulators/anti-TNF $\alpha$  antibodies). The placebo was selected as a comparator for objective evaluation of efficacy and safety.

# 6.2.4 Justification of the Dosage and the Evaluation Period

In the Phase 3 study outside Japan in CD patients (C13007) dosed 300 mg of MLN0002 at Weeks 0, 2, 6 and subsequently every 8 weeks or 4 weeks, similar efficacy was observed in either dosage with no safety issues[9]. The serum MLN0002 concentration was similar inside/outside Japan, and saturation of  $\alpha_4\beta_7$  receptors was observed mostly continuously from the first dose. From the above, the dosage in the study was selected as 300 mg of MLN0002 to be dosed at Weeks 0, 2, 6 and subsequently every 8 weeks in a similar manner as that in C13007 study.

The primary efficacy endpoint in the induction phase will be evaluated at Week 10, since results from the Phase 3 study outside Japan in CD patients (C13011) have suggested that efficacy of the induction therapy is improved at Week 10 than that at Week 6. It has been decided that the

maintenance phase is to start from Week 14, and the primary efficacy endpoint in the maintenance phase will be evaluated at 46 weeks after enrollment into maintenance phase (Week 60) in the similar manner as that in C13007 study.

Meanwhile, non-responders at Week 10 may be enrolled into the open-label cohort for re-induction of the drug and the maintenance therapy, and receive 300 mg of MLN0002 at Weeks 0x, 2x, 6x and subsequently every 8 weeks for 46 weeks (minimum) to 94 weeks (maximum). Subjects who experienced disease worsening or received rescue treatments during the maintenance phase, or those who completed Week 60 of the maintenance phase can be enrolled into the open-label cohort to receive the study drug in the same manner. As safety was demonstrated in the C13007 study when MLN0002 was dosed at Weeks 0, 2 and subsequently every 4 weeks, enrollment into the open-label cohort was judged to impose no safety issues.

The elimination half-life of MLN0002 was 15 to 22 days at the dose of 2 to 10 mg/kg[5]. Additionally, saturation of  $\alpha_4\beta_7$  receptors was durable at the dose of 300 mg for 16 weeks after the last dose, and decreased subsequently over time. The end-of-study examination for safety evaluation after the last dose will be conducted in a similar manner as that in studies outside Japan in all subjects who received the study drugs at 16 weeks after the last dose that is almost  $\geq$ 5-times longer period than the elimination half-life and by which saturation of  $\alpha_4\beta_7$  receptors may be durable.

PML has been reported in subjects who received natalizumab, an  $\alpha_4$  integrin antagonist[12]. MLN0002 is considered unlikely to increase PML risk since it specifically binds to the intestine tropism  $\alpha_4\beta_7$  integrin, and no PML was observed in clinical trials inside/outside Japan so far. However, the number of subjects who received MLN0002 was not large because of the clinical trial stage, and the potential PML risk is difficult to be ruled out. Therefore, the follow-up survey will be performed every 6 months up to 2 years after the last dose of the study drug for evaluation of potential PML risk of the drug.

# **6.2.5** Justification of Endpoints

The CDAI score was used as the disease activity index for CD in C13007 study and C13011 study[9][10]. The CDAI score, extensively used as an efficacy index for evaluation of CD inside/outside Japan, was selected as the evaluation index in the study. The clinical response and clinical remission based on the CDAI score were defined in the same manner as those in C13007 study and C13011 study.

# 6.3 Premature Termination or Suspension of Study or Investigational site

## 6.3.1 Criteria for Premature Termination or Suspension of the Study

The study will be completed as planned unless one or more of the following criteria are satisfied that require temporary suspension or early termination of the study.

- New information or other evaluations regarding the safety or efficacy of the study drug that indicates a change in the known risk/benefit profile for the compound, such that the risk/benefit is no longer acceptable for subjects participating in the study.
- Significant violation of Good Clinical Practice (GCP) that compromises the ability to achieve the primary study objectives or compromises subject safety.

# 6.3.2 Criteria for Premature Termination or Suspension of Investigational Sites

A study site may be terminated prematurely or suspended if the site (including the investigator) is found in significant violation of GCP, protocol, or contractual agreement, is unable to ensure adequate performance of the study, or as otherwise permitted by the contractual agreement.

# 6.3.3 Procedures for Premature Termination or Suspension of the Study or the Participation of Investigational Site(s)

When the sponsor, the IRB or regulatory authorities has decided to suspend or terminate the study or participation of a study site, the sponsor will designate a procedure to be applied in the study. The study site should follow the designated procedures to suspend or terminate the study.

# 7.0 SELECTION AND DISCONTINUATION/WITHDRAWAL OF SUBJECTS

All inclusion/exclusion criteria including test results must be confirmed prior to enrollment into the induction phase.

## 7.1 Inclusion Criteria

Subject eligibility is determined according to the following criteria:

- 1. In the opinion of the investigator, a subject is capable of understanding and complying with protocol requirements.
- 2. A subject who is capable of entering the signature and the date on the informed consent by himself/herself or by the subject's legally acceptable representative, if applicable, prior to initiation of study procedures.
- 3. A subject aged 15 to 80 (inclusive) at the time of signing the informed consent (regardless of sexes).
- 4. A male subject, who has no sterilization history and whose female partner has child-bearing potential, who agreed with taking proper contraception during the period from the time of signing on the informed consent form through 6 months after the last dose of the study drug.
- 5. A female subject with child-bearing potential (having no history of sterilization or whose last menstruation was within 2 years) whose male partner is not receiving contraceptive treatment, and agreed to take proper contraception during the period from the time of signing on the informed consent form through 6 months after the last dose of the study drug.
- 6. Subjects with a diagnosis of the small intestine type, the large intestine type or the small/large intestine type of CD based on the Revised Diagnostic Criteria for Crohn's Disease issued by "Research Group for Intractable Inflammatory Bowel Disease" Designated as Specified Disease by the MHLW of Japan (2012) (see Appendix C) at least 3 months before the start of administration of study drug.
- 7. Subjects with the CDAI score of 220≤ and ≤450 points at the first dose of the study drug, and also meeting any of the following:
  - Subjects with a CRP level of >0.30 mg/dL at the screening test.
  - Subjects confirmed to have irregular-to-round shaped ulcers or multiple aphtha in the small or large intestine extensively (≥10 lesions) in the endoscopy or the imaging test within 4 month before the first dose of the study drug.
  - Subjects confirmed to have longitudinal ulcers or a cobblestone appearance in the small or large intestine in the endoscopy or the imaging test within 4 months before the first dose of the study drug.
- 8. Subjects whose complication of colon cancer or dysplasia had to be ruled out by total colonoscopy at the start of the study drug administration (or the results from total colonoscopy performed within 1 year before giving consent are available), if subjects met any of the

followings; subjects with extensive or limited colitis of  $\geq 8$  years duration, subjects aged  $\geq 50$  years, or subjects with a first-degree family history of colon cancer.

9. Subjects meeting the following treatment failure criteria with at least one of the following agents within 5 years before the time of signing on the informed consent form:

## Corticosteroids

- Resistance: subjects whose response was inadequate after treatment of  $\geq$ 40 mg/day for  $\geq$ 1 week <sup>3</sup>(oral or IV) or 30 to 40 mg/day for  $\geq$ 2 weeks (oral or IV).
- Dependence: subjects for which it is difficult to reduce the dosage to <10 mg/day due to recurrence during gradual dose reduction (oral or IV).
- Intolerance: subjects who were unable to receive continuous treatment due to adverse reactions (e.g., Cushing's syndrome, osteopenia/osteoporosis, hyperglycaemia, insomnia, infection).

# • Immunomodulators (AZA, 6-MP or MTX)

- Refractory: subjects whose response was inadequate after treatment for  $\ge$ 12 weeks.
- Intolerance: subjects who were unable to receive continuous treatment due to adverse reactions (e.g., nausea/vomiting, abdominal pain, pancreatitis, LFT abnormalities, lymphopenia, TPMT genetic mutation, infection).

## • Anti-TNFα antibodies

- Inadequate response: subjects whose response was inadequate after the induction therapy in the dosage described in the package insert.
- Loss of response: subjects who had recurrence during the scheduled maintenance therapy after achievement of clinical response (those who withdrew for other reasons than relapse are not applicable here).
- Intolerance: subjects who were unable to receive continuous treatment due to adverse reactions (e.g., infusion-related reaction, demyelination disease, congestive heart failure, infection).

# 7.2 Exclusion Criteria

Subjects meeting any of the following criteria will not be eligible in the study:

- 1. Subjects having or suspected to have abdominal abscess.
- 2. Subjects with a history of subtotal or total colectomy.
- 3. Subjects with a history of  $\geq 3$  enterectomy, or a history of diagnosis of short bowel syndrome.
- 4. Subjects with ileostomy, colostomy, internal fistula or severe intestinal stenosis.

<sup>&</sup>lt;sup>3</sup>The dosages of corticosteroids represent, hereafter, the converted dosage of prednisolone.

- 5. Subjects having a treatment history with natalizumab, efalizumab or rituximab.
- 6. Subjects who started oral 5-ASA, probiotics, antibiotics for CD treatment, or oral corticosteroids (≤30 mg/day) within 13 days before the first dose of the study drug. Subjects who have used these drugs for at least 14 days before the first dose of the study drug, and who changed dosage of or discontinued these drugs within 13 days before the first dose of the study drug.
- 7. Subjects who have received 5-ASA, corticosteroid enemas/suppositories, corticosteroid IV infusion, oral corticosteroid at >30 mg/day, drugs for diarrhea-predominant irritable bowel syndrome, or Chinese herbal medicine for the CD treatment (e.g., Daikenchuto) within 13 days before the first dose of the study drug.
- 8. Subjects who have received AZA, 6-MP or MTX within 27 days before the first dose of the study drug However, this will not apply to subjects who have used these drugs for 83 or more days before the first dose of the study drug and continued the steady dose administration of the drugs for 27 or more days before the first dose of the study drug.
- 9. Subjects who have received cyclosporine, tacrolimus, tofacitinib or any study drugs of low-molecular compound for CD treatment within 27 days before the first dose of the study drug.
- 10. Subjects who have received adalimumab within 27 days before the first dose of the study drug or any biologic agents other than adalimumab within 55 days before the first dose of the study drug. However, this will not apply to subjects who have topically received these drugs (e.g., intraocular injection for treatment of age-related macular degeneration).
- 11. Subjects who have received any live-vaccinations within 27 days before the first dose of the study drug.
- 12. Subjects who underwent the enterectomy within 27 days before the first dose of the study drug or those anticipated to require an enterectomy during the study.
- 13. Subjects who have received leukocytapheresis or granulocyte apheresis within 27 days before the first dose of the study drug.
- 14. Subjects who received central venous nutrition therapy or enteral total nutrition therapy, or fasted within 20 days before the first dose of the study drug.
- 15. Subjects who received an enteral nutrient of >900 kcal/day or who will begin to receive an enteral nutrient of ≤900 kcal/day within 20 days before the first dose of the study drug. Subjects who had received an enteral nutrient of ≤900 kcal/day earlier than 21 days before the first dose of the study drug, and modified or discontinued the dosage within 20 days before the first dose of the study drug.
- 16. Subjects who have been infected with an intestinal pathogen including clostridium difficile or cytomegalovirus within 27 days before the first dose of the study drug.

- 17. Subjects with evidence of adenomatous colonic polyps that need to be removed at the start of study drug administration.
- 18. Subjects with a history or a complication of large or small intestinal dysplasia.
- 19. Subjects suspected to have enteritis other than CD.
- 20. Subjects indicated in the screening test as HBs antigen-positive or HCV antibody-positive Subjects indicated as HBc antibody-positive or HBs antibody positive even though HBs antigen-negative However, the criteria will not apply to those with only HBs antibody-positive due to HBV vaccination, HBV-DNA-negative, HCV antigen-negative or HCV-RNA-negative.
- 21. Subjects who have or are suspected to have a history of tuberculosis (including those whose findings in the chest imaging procedure at screening showing anamnesis of tuberculosis) However, the criteria will not apply to those who had completed prophylactic treatment with isoniazid, and who have been receiving prophylactic isoniazid for 21 days or longer before the first dose of the study drug (the latter may initiate study drug administration with screening phase extended to 28 days at maximum for prophylactic treatment to become 21 days or more).
- 22. Subjects indicated as positive in T-SPOT or QuantiFERON at screening test.
- 23. Subjects who have a history or complication of congenital or acquired immunodeficiency syndrome (e.g., not-classifiable immunodeficiency, HIV infection or organ transplantation).
- 24. Subjects who were affected by extraintestinal infection (e.g., pneumonia, sepsis, active hepatitis or pyelonephritis) within 27 days before the first dose of the study drug.
- 25. Subjects who have treatment history with MLN0002.
- 26. Nursing mothers during the screening phase, or female subjects indicated positive in urine pregnancy test either at the screening or baseline.
- 27. Subjects having serious complications in the heart, lung, liver, kidney, metabolism, gastrointestinal system, urinary system, endocrine system or blood.
- 28. Subjects with a history of an operation requiring general anesthesia within 27 days before the first dose of the study drug, or with a schedule of an operation requiring hospitalization during the study period.
- 29. Subjects having a complication or a history of malignancy However, it will not apply to the following subjects;
  - Subjects who had a curative resection of localized skin basal cell carcinoma or had completed curative radiotherapy.
  - Subjects who have not experienced recurrence for 1 year or longer since completion of curative resection or curative radiotherapy for skin squamous cell carcinoma.

• Subjects who have not experienced recurrence for 3 years or longer since completion of curative resection or curative radiotherapy for intraepithelial carcinoma of uterine cervix.

For subjects having a substantially distant history of malignancy (e.g., 10 years or longer without recurrence since treatment completion), the Investigator and the sponsor will discuss to decide eligibility on the basis of type of malignancy and treatment applied.

- 30. Subjects having a history or a complication of the central nervous disorder, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
- 31. Subjects for which any subjective symptoms in the Subjective PML checklist were found at the screening or baseline.
- 32. Subjects for which any of the following laboratory abnormalities were found at the screening;

• Hemoglobin ≤8 g/dL

• White blood cells  $\leq 3,000/\mu L$ 

• Lymphocytes  $\leq 500/\mu L$ 

• Platelets  $\leq 100,000/\mu L$ , or  $\geq 1,200,000/\mu L$ 

• ALT and AST  $\geq 3 \times \text{upper limit of normal (ULN)}$ 

• ALP ≥3×ULN

• Creatinine  $\geq 2 \times ULN$ 

- 33. Subjects having a history or a complication of alcohol dependence or illicit drug use within one year before the first dose of the study drug.
- 34. Subjects having a history or a complication of psychotic disorder that may obstruct compliance with the study procedures.

## 7.3 Excluded Medications and Treatments

Excluded medications and treatments are listed in Table 7.a. However, some of the drugs may be used concurrently under the conditions provided in the table. Subjects will be instructed not to take any drugs, including over-the-counter products (OTCs), without first consulting with the investigator.

Table 7.a List of Excluded Drugs and Treatments

| | Prohibited Period <sup>1)</sup> | | | Conditions in Concurrent Use | |
|---|---|---|---|---|---|
| Drugs/Treatment | | | | Screening Phase/<br>Induction Phase/Maintenance Phase | Open-label<br>Cohort |
| Oral 5-ASA Probiotics <sup>2)</sup> Antibiotics for CD treatment | Day -13 | _ | the last dose | at the same dosage from Day-13. Dose reduction | Allowed to<br>be used<br>(without<br>limitation) |
| Oral corticosteroids (≤30 mg/day) | Day -13 | - | 16 weeks after | Should be initiated before Day-14 and | Same as on |

| | | Conditions in Concurrent Use |
|---|---|---|
| Drugs/Treatment | Prohibited Period 1) | Screening Phase/ Open-label Induction Phase/Maintenance Phase Cohort |
| | the last d | ose continued at the same dosage from Day-13. the left As per the Dose Reduction Schedule for corticosteroids (see Section 7.3.2). |
| 5-ASA enemas<br>5-ASA suppositories | Day -13 - 16 weeks the last d | |
| Corticosteroid enemas<br>Corticosteroid suppositories<br>(including corticosteroid pretreatment<br>prior to endoscopy) | Day -13 - 16 weeks the last d | |
| Corticosteroid IV infusion | Day -13 - 16 weeks at the last d | |
| Oral corticosteroids (>30 mg/day) | Day -13 - 16 weeks at the last d | |
| Therapeutic drugs for diarrhea-predominant irritable bowel syndrome | Day -13 - 16 weeks the last d | |
| Chinese herbal medicines for UC treatment (eg, Daikenchuto) | Day -13 - 16 weeks the last d | |
| AZA<br>6-MP<br>MTX | Day -27 – 16 weeks the last d | |
| Tacrolimus Cyclosporine Tofacitinib | Day -27 – 16 weeks the last d | |
| Study drugs of low-molecular compounds for CD treatment | Day -27 – 16 weeks the last d | |
| Adalimumab | Day -27 - 16 weeks the last d | |
| Natalizumab<br>Efalizumab<br>Rituximab<br>MLN0002 | (previous) - 16 weeks the last d | |
| Other biologics than the above (including infliximab. Topical use was allowed) | Day -55 - 16 weeks the last d | |
| Live-vaccinations | Day -27 – 6 months a | |
| Enterectomy [Other surgical treatments than the enterectomy including (treatment-emergent) abscess drainage or the Seton method for the anal lesion may be performed] | Day -27 – 16 weeks the last d | |
| Leukocytapheresis or granulocyte apheresis | Day -27 – 16 weeks the last d | |

| Drugs/Treatment | Prohibited Period 1) | | Conditions in Concurrent Use | |
|---|---|---|---|---|
| | | | Screening Phase/<br>Induction Phase/Maintenance Phase | Open-label<br>Cohort |
| Central venous nutrition therapy<br>Enteral total nutrition therapy<br>Fasting | Day -20 – | 16 weeks after<br>the last dose | | _ |
| Enteral nutrients (>900 kcal/day) | Day -20 – | 16 weeks after<br>the last dose | _ | _ |
| Enteral nutrients (≤900 kcal/day) | Day -20 – | 16 weeks after<br>the last dose | Should be initiated before Day-21 and continued at the same dosage from Day-20. The dosage may be modified after Week 10, however it should preferably remain the stable dose and not exceed the initial dosage at the first dose of the study drug. | left |
| Surgeries requiring general anesthesia | Day -27 – | 16 weeks after<br>the last dose | _ | _ |

<sup>1)</sup> Day 1 is defined as the date of the first dose of the study drug and Day -1 is defined as the day before the Day 1 for calculation.

## 7.3.1 Rescue Treatments

Drugs or treatments not permitted in Table 7.a may be used as rescue treatments (see Section 3.1 for the definition) only in urgent cases such as worsening of CD otherwise safety of the subject is judged not to be secured.

The subjects who received any rescue treatments in the induction phase should withdraw from the study. The subjects who received any rescue treatments in the maintenance phase should discontinue the maintenance phase and may be enrolled into the open-label cohort, however withdrawal should be considered in the subjects intending to receive any unavailable treatment in the open-label cohort. For the subjects who received any rescue treatments in the open-label cohort, withdrawal should be considered (see Section 7.5).

## 7.3.2 Dose Reduction Schedule of Corticosteroids

Dosage of a corticosteroid, if used concurrently, should not be modified until Week 10 after the first dose of the study drug in principle. When the CDAI-70 response (see Section 3.1 for the definition) was achieved at Week 10 or later, the dose reduction of the corticosteroid will be initiated as per the following schedule from the visit when the CDAI-70 response was observed, where possible.

## Dose Reduction Schedule:

- When >10 mg/day was dosed, the dosage will be gradually reduced by 5 to 10 mg/2 weeks to reach 10 mg/day
- When ≤10 mg/day was dosed or achieved by gradual reduction, the dosage will be gradually reduced by 2.5 to 5 mg/2 weeks to achieve corticosteroid-free

<sup>2)</sup> Such as VSL#3. The bifidobacterium preparation or any foods are not applicable.
When dose reduction is required earlier than Week 10 due to adverse reactions of the corticosteroid, only small doses of not more than 5 mg/2 weeks should be gradually reduced.

When any symptoms recur with the dose reduction of the corticosteroid, the dosage may be increased up to the initial dose (it will not apply to rescue treatments). Subsequently, when clinical response was observed again, the dose reduction will be initiated preferably as per the above schedule from the visit when the clinical response was observed.

Of note, higher dosage than the initial dosage, if used for recurrence, will be considered as a rescue treatment (see Section 7.3.1 for rescue treatments).

## 7.4 Subject Management

- 1. Subjects should be instructed to be sure to see the physician and take specified examinations at the specified date and time. In addition, subjects should be instructed to inform the investigator or the sponsor immediately in the case that they cannot visit.
- 2. Subjects should be instructed to make entries in the subject's diary throughout the period from the time of signing on the informed consent form to the last dose of the study drug and to bring the diary with them at each visit.
- 3. Subjects should be instructed to preferably visit under fasted condition at visits for blood biochemistry test.
- 4. Subjects should be instructed to report any worsening of symptoms that occurred at any time other than visits, if any, to the investigator or the sponsor via telephone or the like to seek instructions.
- 5. Subjects should be instructed to report details, onset date, intensity, outcome and outcome date of subjective symptoms/objective findings to the investigator during their visit.
- 6. Subjects should be instructed to report course and details of the treatment to the investigator if they visited other medical institutions during the period from the time of signing on the informed consent form to 16 weeks after the last dose of the study drug.
- 7. Subjects should be instructed to inform a physician in a medical institution of his/her participation in the study, if he/she visited other medical institutions during the period from the time of signing on the informed consent form to 16 weeks after the last dose of the study drug.
- 8. Subjects should be instructed not to use any drugs including OTCs other than drugs instructed by the investigator without prior consultation (except urgent cases).
- 9. Male subjects without a sterilization history and whose female partner has child-bearing potential should be instructed to take proper contraception during the period from the time of signing on the informed consent form to 6 months after the last dose of the study drugs.

- 10. Female subjects with child-bearing potential whose male partner has no sterilization history should be instructed to take proper contraception during the period from the time of signing on the informed consent form to 6 months after the last dose of the study drugs.
- 11. Subjects should be instructed to avoid surfeit, extreme changes in diet, excessive exercise/action throughout the period from the time of signing on the informed consent form to the last dose of the study drug. Subjects should be instructed in an especially careful manner because treatment-emergent change of symptoms may lead to changes in diet.
- 12. Subjects should be instructed not to donate their blood during the period from the time of signing on the informed consent form to 6 months after the last dose of the study drug.
- 13. Subjects should be instructed to report any feelings of infusion reaction (e.g., rash, pruritus, flushing or urticaria) to the investigator immediately.

## 7.5 Criteria for Discontinuation or Withdrawal of a Subject

The primary reason for discontinuation or withdrawal of a subject from the study should be recorded in the case report form ([e]CRF) using the following categories. See Section 9.1.21 for subjects who withdrew during the screening phase.

#### 1. Pretreatment Events or AEs

The subject has experienced a PTE or AE that requires early termination because continued participation imposes an unacceptable risk to the subject's health or the subject is unwilling to continue because of the PTE or AE.

- Liver Function Test Abnormalities
  Discontinuation of the study drug should be considered with appropriate clinical follow-up (including repeat laboratory tests, until a subject's laboratory profile has
  - returned to normal/baseline status, see Section 9.1.12), if the following circumstances occur at any time during study drug treatment:
  - ALT or AST  $>8\times$ ULN, or
  - ALT or AST >5×ULN and persists for more than 2 weeks, or
  - ALT or AST >3×ULN in conjunction with elevated total bilirubin >2×ULN or international normalized ratio (INR) >1.5, or
  - ALT or AST >3×ULN with appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia.

#### 2. Major protocol deviation

The discovery post-randomization in the induction phase that the subject failed to meet protocol inclusion criteria or did not adhere to protocol requirements, and continued participation poses an unacceptable risk to the subject's health.

Note: The visit for evaluation of the primary efficacy endpoint in the induction phase (Visit 5), when notably deviated beyond the acceptable window (≥±15 days), should be considered as a major protocol deviation.

#### 3. Lost to follow-up

The subject did not return to the clinic and attempts to contact the subject were unsuccessful. Attempts to contact the subject must be documented.

### 4. Voluntary withdrawal.

The subject wishes to withdraw from the study. The reason for withdrawal, if provided, should be recorded in the (e)CRF.

Note: All attempts should be made to determine the underlying reason for the withdrawal and, where possible, the primary underlying reason should be recorded (i.e., withdrawal due to an AE or lack of efficacy should not be recorded in the "voluntary withdrawal" category).

#### 5. Study termination

The sponsor, the IRB or regulatory authorities decided to terminate the study.

#### 6. Pregnancy

The subject is found to be pregnant.

Note: If the subject is found to be pregnant, the subject must be withdrawn immediately. The procedure is described in Section 9.1.13.

#### 7. Lack of efficacy

The investigator has determined that the subject is not benefiting from investigational treatment; and, continued participation would pose an unacceptable risk to the subject.

Note: A subject who received any rescue treatments due to lack of efficacy in the induction phase should withdraw from the study immediately. For a subject who received any rescue treatments in the open-label cohort, and meets criteria for the sustained non-response or the disease worsening, withdrawal due to lack of efficacy will be considered

#### 8. Other

Note: The specific reasons should be recorded in the "specify" field of the (e)CRF.

#### 7.6 Procedures for Discontinuation or Withdrawal of a Subject

The investigator may terminate a subject's study participation at any time during the study when the subject meets the study termination criteria described in Section 7.5. In addition, a subject may discontinue his or her participation without giving a reason at any time during the study. Should a subject's participation be discontinued, the primary criterion for termination must be recorded. In addition, efforts should be made to perform all procedures scheduled for the early termination visit.

#### 8.0 CLINICAL STUDY MATERIAL MANAGEMENT

This section contains information regarding all drugs and materials provided directly by the sponsor, and/or by other means, that are required by the study protocol, including important sections describing the management of clinical trial materials.

## 8.1 Study Medication and Materials

## 8.1.1 Dosage Form, Manufacturing, Packaging, and Labeling

## 8.1.1.1 Study Drug

In this protocol, the term of study drugs refers to all or any of the drugs defined below.

Table 8.a Study drug

| Name of the study<br>drugs | Chemical name of active ingredients (Nonproprietary names) | Formulations | Contents |
|---|---|---|---|
| MLN0002<br>300 mg for infusion | Human IgG <sub>1</sub> monoclonal antibody [vedolizumab (INN)] against human $\alpha_4\beta_7$ integrin | Parenteral solution | Contains 300 mg* of MLN0002 in one vial |
| Placebo for infusion | Not applicable | _ | Empty |

<sup>\*</sup>lyophilized preparation

Appearance is identical among vials of the study drugs. Each vial will be labeled to be packed into the outer package. The outer package will be labeled with the statement that contents are study drugs, the name of the study drug, quantity, the name and address of the sponsor, the serial number, the storage and the expiration date. Examples of labels on vials or outer packages are shown in the Figure 8.a and Figure 8.b, respectively. Of note, the serial numbers and expiration dates of the study drugs should be in accordance with the separately specified written procedure.

Figure 8.a Labels on Vials

MLN0002/CCT-001

MLN0002 (300 mg) for infusion

Serial number: Z ......

MLN0002/CCT-001

NOT for infusion to subjects

For vials of MLN0002 (300 mg)

For vials of placebo

Figure 8.b A Label on Outer Packages

| Study drug 1 vial | |
|---|---|
| MLN0002 DB for infusion MLN0002/CCT-001 Drug number: | Serial number: DB<br>Expiration date:See the procedure for<br>study drug control<br>Storage: refrigerated (2 to 8 °C) |
| Subject Identification Code: | Note The outer package should be kept to be collected by the Sponsor. |
| Timing for infusion: | Takeda Pharmaceutical Company<br>Limited |
| Week | 1-1, Doshomachi 4-chome, Chuo-ku,<br>Osaka-shi |

## 8.1.1.2 Materials

The following materials will be used at the time of infusion of the study drugs in principle. However, the material control should be in accordance with the separately specified written procedures.

**Table 8.b** Materials

| Intended use | Materials | Examples |
|---|---|---|
| Preparation of<br>study drugs | A syringe for preparation | A 5 or 10 cc latex-free syringe |
| | Water for injection | Water for injection in a container with volume of 10 mL or larger |
| | An injection needle for preparation | An injection needle of 18G stainless steel |
| | Physiological saline | Sterilized 100 mL (specification) 0.9% NaCl solution |
| Infusion of<br>study drugs | An IV infusion kit | An IV infusion kit to set the injection site beneath an infusion tube |
| | An injection needle for infusion | A winged needle for IV infusion |
| | Physiological saline<br>(for priming/flushing IV<br>infusion lines) | Sterilized 50, 100 or 250 mL (specification) 0.9%<br>NaCl solution |

## 8.1.2 Storage

Temperature during storage should be refrigerated (2 to 8°C). However, it may be deviated temporally (for 7 days) in the range from -70 to 40°C.

All study drugs must be kept in an appropriate, limited-access, secure place until used or returned to the sponsor or its designee for destruction. All sponsor-supplied study drugs must be stored under the conditions specified on the label, and remain in the original container until dispensed. A daily temperature of the study drug storage area must be determined and recorded every working day.

#### 8.1.3 Dose and Regimen

Table 8.c Dose and Regimen

| Study Drugs | Preparation and Regimen |
|---|---|
| Placebo for infusion | Add 5 mL of water for injection to approximately 100 mL of saline and infuse intravenously over 30 minutes*. |
| MLN0002 (300 mg) for infusion | One vial of MLN0002 (300 mg) for infusion is reconstituted in 4.8 mL of water for injection. Add 5.0 mL of the solution to approximately 100 mL of saline for dilution and infuse intravenously over 30 minutes*. |

<sup>\*</sup>May be infused over 60 minutes at maximum.

Study drug preparators should prepare study drugs. A study drug preparators should not be an evaluator throughout induction and maintenance phases. Study drug preparators will prepare study drugs in line with the drug numbers prescribed by the investigator or his/her designee. The details of the study drug preparation method should be in accordance with the separately specified written procedure.

Serious infusion reaction should be treated properly, if any, e.g., immediate use of epinephrine and parenteral diphenhydramine.

#### 8.1.4 Overdose

Overdose is defined as a known deliberate or accidental administration of a study drug at a dose above the specification in the study protocol.

All cases of overdose (with or without associated AEs) will be documented on an Overdose page of the (e)CRF, in order to capture this important safety information consistently in the database. AEs associated with an overdose will be documented on AE (e)CRF(s) according to Section 10.0, PTEs and AEs.

SAEs associated with overdose should be reported in accordance with the procedure specified in Section 10.2.2 Collection and Reporting of SAEs.

Subjects overdosed should be treated by the investigator based on symptoms.

## 8.2 Procedures for Allocation, Prescription and Infusion of Study Drugs

A study drug number will not be identical at each time. For allocation of subjects to study drugs, Investigators or his/her designee will access the website of the registration center at each visit for infusion to obtain a study drug number from the registration center. Investigators or his/her designee will prescribe the study based on the obtained study drug number. The study drug number should be recorded in (e)CRF at each administration visit.

Details for using the website of the registration center will be in accordance with the separately specified written procedures.

## 8.3 Preparation and Retention of the Allocation Table

A person in charge of allocation (appointed by the sponsor) will prepare the allocation table. Information of allocation should be kept in a secure place with limited access by unauthorized people.

#### 8.4 Preservation of Blindness

The emergency key will be kept in the emergency key control center until emergent key-breaking or completion of database lock of all subjects.

In the study, allocations must not be disclosed to any person until opening of the study drug allocation table, while the study drug preparators may be aware of allocations in the course of study drug preparation.

Furthermore, test results of serum drug concentration and HAHA/neutralizing antibody may be an obstacle in preservation of blindness in the study, therefore these final test results should be kept undisclosed outside in the test laboratory until opening of the study drug allocation table, and will be reported to the investigator through the sponsor upon opening. However, if a test result must be disclosed before opening, the test result may be reported to the sponsor or the like after necessary actions taken to preserve blindness (e.g., renumbering of study drugs), so that persons in charge in the test laboratory would be unable to identify subjects. Detailed procedures should be in accordance with the separately specified written procedure.

#### 8.5 Procedures for Blind-Breaking

The study drug blind will not be broken by the investigator unless information concerning the study drug is necessary for the medical treatment of the subject.

In blind-breaking, the investigator may obtain study drug allocation information from the emergency key control center (see the Annex for contacts).

In blind-breaking, the investigator will enter the date/time and rationale of the blind-breaking on the record of emergency key opening to be submitted to the sponsor. The same information (except time) will be recorded on (e)CRF.

If any site personnel is unblinded, the study drug must be stopped immediately and the subject must be withdrawn from the study.

## 8.6 Control and Disposal of Sponsor-Supplied Drugs

The Study Drug Administrator will receive the written procedure prepared by the sponsor relating to handling, storing and controlling study drugs to properly control sponsor-supplied study drugs and materials in accordance with the written procedure. Similarly, the investigator will receive the same written procedures from the sponsor. The written procedure describes procedures to ensure proper receipt, handling, storing, controlling and prescription of the sponsor-provided study drugs and materials, as well as return of unused study drugs and materials to the sponsor or other disposition.

The Study Drug Administrator will return unused study drugs and materials to the sponsor immediately after study completion in the study site.

#### 9.0 STUDY PLAN

#### 9.1 Study Procedures

The following sections describe the study procedures and data to be collected. For each procedure, subjects should be assessed by the same investigator or site personnel, where possible. The Study schedule is provided in Appendix A.

#### 9.1.1 Informed Consent Procedure

The requirements of the informed consent are described in Section 15.2.

The informed consent must be obtained prior to the subject entering into the study, and before any protocol-directed procedures are performed.

Dosage of prior therapeutic drugs will be modified or discontinued for the study enrollment, if needed, after acquisition of the informed consent for participation in the study.

Subject Identification Code will be provided for each subjects at the time of explanation of the informed consent, and used throughout the study.

### **Pharmacogenomic Informed Consent Procedure**

A separate informed consent form pertaining to storage and banking of the sample must be obtained prior to collecting a blood sample for Pharmacogenomic Research for this study. The provision of consent to collect and analyze the pharmacogenomic sample is independent of consent to the other aspects of the study.

## 9.1.2 Demographics, Medical History, and Medication History Procedure

As demographic data, dates of birth, sex and smoking histories will be obtained. In addition, the following CD-related items will be obtained.

- Date Primary Disease Diagnosed
- The following item as defined in the Revised Diagnostic Criteria for CD (Appendix C) issued by "Research Group for Intractable Inflammatory Bowel Disease" Designated as Specified Disease by the MHLW of Japan (2012)
  - Disease localization by extent of the CD lesions (small-intestinal, large-intestinal or small/large-intestinal)
- History of treatment failure with the following drugs within 5 years before acquisition of the informed consent
  - Corticosteroids (resistance/dependence/intolerance)
  - Immunomodulators (AZA, 6-MP or MTX) (refractory/intolerance)
  - Anti-TNFα antibodies\* (inadequate response/loss of response/intolerance)

\* For inadequate response and loss of response, the name and the first and last administration dates of the drug will be recorded as well. For intolerance, the name of the drug and the side-effect leading to discontinuation will be recorded as well.

For disease histories, any clinically relevant diseases or symptoms will be obtained, which were judged as disease histories in evaluation in the study by a physician, including extra-intestinal manifestations, pouchitis, infectious enteritis, toxic megacolon, stenosis, fistula that has recovered/resolved within 1 year before acquisition of the informed consent. In addition, any previous malignancies and enterectomy for CD will be obtained. Ongoing conditions or diseases are considered as concurrent medical conditions (see Section 9.1.7).

For prior therapeutic drugs, all of the following will be obtained.

- Biological drugs for CD treatment discontinued before acquisition of the informed consent.
- Low-molecular compounds for CD treatment discontinued within 4 weeks before acquisition of the informed consent.

Of note, agents applied for procedures including endoscopy will not be considered as prior therapeutic drugs and also not be documented in the (e)CRF.

#### 9.1.3 Physical Examination Procedure

Physical examination in the following body sites will be performed before study drug administration if it is the day of study drug administration.

- (1) eyes, (2) ears, nose, throat, (3) cardiovascular system, (4) respiratory system,
- (5) gastrointestinal system, (6) dermatologic system, (7) extremities, (8) musculoskeletal system,
- (9) nervous system, (10) lymph nodes, and (11) other. During infusion and 1 hour after infusion of the study drug, infusion reactions (e.g., rash, pruritus, flushing or urticaria) will be observed, and clinically relevant abnormalities will be assessed as compared to physical examination results performed before study drug administration.

#### 9.1.4 Weight, Height and BMI

Body weight and height will be measured before administration of the study drug if it is the day of study drug administration. In addition, BMI will be calculated by the sponsor with the following formula;

Metric: BMI = weight  $(kg)/[height (m)]^2$ 

Height will be collected in centimeters without decimal places and weight will be collected in kilograms to 1 decimal place, results for BMI will be expressed with 1 decimal place.

#### 9.1.5 Vital Sign Procedure

As vital signs, body temperature (axilla), blood pressure while sitting (rest for 5 minutes or longer), and pulse (bpm) will be measured before administration of the study drug if it is the day of study drug administration.

## 9.1.6 Documentation of Concomitant Medications and Non-drug Therapy

Concomitant medication is any drug given in addition to the study medication. These may be prescribed by a physician or obtained by the subject over the counter. Concomitant medication is not provided by Takeda. At each study visit, subjects will be asked whether they have taken any drug other than the study drug (used from the time of signing on the informed consent form through the end-of-study examination), and all drugs including vitamin supplements, OTC drugs, and oral herbal preparations, must be recorded in the (e)CRF. In addition, for concomitant drugs for CD treatment, class of the concomitant drug (5-ASA, corticosteroids, immunomodulators, enteral nutrition, or others), and applicability to a rescue treatment will be recorded in the (e)CRF.

Concomitant treatments are defined as any treatments for CD other than pharmacotherapy, including enterectomy and other surgical treatments (e.g., abscess drainage or the seton method for the anal lesion). All concomitant treatments that were conducted during the period from acquisition of the informed consent until the end-of-study examination will be obtained. Additionally, applicability of the concomitant treatment to a rescue treatment will be recorded in the (e)CRF.

Of note, agents applied for test procedures including endoscopy will not be considered as concomitant drugs and will also not be documented in the (e)CRF.

#### 9.1.7 Documentation of Concurrent Medical Conditions

Concurrent medical conditions are those significant ongoing conditions or diseases that are present at the time of signing on the informed consent form. This includes clinically significant laboratory, ECG, or physical examination abnormalities noted at screening/baseline examination. The condition (i.e., diagnosis) should be described. In addition, CD-related extra-intestinal manifestations will be recorded in the (e)CRF.

#### 9.1.8 The Patient Diary

The patient diaries are used for calculation of the CDAI scores. At each visit, patient diaries to be entered from the visit to the next visit will be handed to subjects. A subject will be instructed to record the following items in the diary and bring it at the next visit.

- Number of liquid or very soft stools
- Scores of abdominal pain
- Scores of general well being
- Fever of ≥37.8°C
- Use of antidiarrheal drugs or opiates

Contents of the patient diaries will be confirmed at each visit. The subject will be asked about omissions or inconsistencies for correction, if any. The patient diaries will be collected to be retained after final confirmation of the contents.

#### 9.1.9 CDAI Score

CDAI scores will be calculated as total scores of the following 8 subscores in the Table 9.a. The necessary information should be entered on the website of the Registration Center for calculation of a CDAI score.

Table 9.a CDAI Scoring System for the Assessment of CD Activity [13]

| (1) Number of liquid or very soft stools | x 2 |
|---|---|
| 7-day total number of liquid or very soft stools (reported on the 7 days immediately prior to the study visit) | |
| (2) Abdominal pain | x 5 |
| 7-day total of daily abdominal pain scores on a 3-point scale: 0=none, 1=mild, 2=moderate, 3=severe (reported on the 7 days immediately prior to the study visit) | |
| (3) General well being | x 7 |
| 7-day total of daily general well-being scores on a 4-point scale: 0=generally well, 1=slightly under par, 2=poor, 3=very poor, 4=terrible (reported on the 7 days immediately prior to the study visit) | |
| (4) Extraintestinal manifestations of CD | x 20 |
| Total number of checked boxes (check all that apply): | |
| □ Arthritis/arthralgia | |
| <ul> <li>□ Iritis/uveitis</li> <li>□ Erythema nodosum/pyoderma gangrenosum/aphthous stomatitis</li> </ul> | |
| ☐ Anal fissure, anal fistula or perianal abscess | |
| □ Other fistula | |
| □ Fever over 37.8°C during the last week | |
| (5) Lomotil/Imodium/opiates for diarrhea | x 30 |
| Yes = 1, No = 0 | |
| (6) Abdominal mass | x 10 |
| None = $0$ , Questionable = $2$ , Definite = $5$ | |
| (7) Hematocrit (%) 1) | x 6 |
| Males: subtract value from 47, Females: subtract value from 42 | |
| (8) Body weight <sup>2)</sup> | x 1 |
| (1 – (Body weight/ Standard Weight)) × 100 | |
| | - |

Contents in the patient diary during the last 10 days before evaluation will be entered on the website of the registration center with regard to each subscore of number of liquid or very soft stools, abdominal pain, general well being, and use of an antidiarrheal drug or an opiate for diarrhea, as well as emergence of fever of ≥37.8°C during the last 1 week. Each subscore will be calculated automatically based on the patient diary during the last 7 days before evaluation except the following days.

- The day of pretreatment for endoscopy
- The day of endoscopy and the next day


Of note, for baseline evaluation (Visit 2), contents of the patient diary during at least 7 days except the above exception days should be entered on the website of the registration center for calculation of CDAI score. The subject visit will be adjusted to have the necessary number of days in the patient diary.

## 9.1.9.1 Calculation of Hematocrit (Ht) level scores

The venous blood will be sampled for determination of Ht level for calculation of the CDAI score.

At baseline (Visit 2), Ht level will be determined in each site on the evaluation day for calculation of the CDAI score, on which eligibility of the subject will be judged prior to initiation of the study drug. The above CDAI score will be the baseline score. If Ht level on the evaluation day is impossible to be obtained, instead Ht level determined during the period from 14 days before evaluation to the evaluation day may be used.

At evaluation of the primary efficacy endpoint (Visit 5), Ht level will be determined in each site on the evaluation day for calculation of the CDAI score, on which clinical response/no-response will be judged in comparison with the baseline score. If Ht level on the evaluation day is impossible to be obtained, instead Ht level determined during the period from 14 days before evaluation to the evaluation day may be used.

At all evaluation except the above, Ht level will be determined in each site on the evaluation day for calculation of the CDAI score, where possible, on which clinical response/no-response will be judged in comparison with the baseline score. If Ht level on the evaluation day is impossible to be obtained, the latest Ht level may be used.

Of note, Ht level for analyses should be determined in the Laboratory Site.

#### 9.1.10 Inflammatory Bowel Disease Questionnaire (IBDQ)

The IBDQ, as composed of a total of 32 questions (each has 1 to 7 points) including abdominal symptoms (10 items), general condition (5 items), emotion (12 items) and social function (5 items), will be calculated as the total scores, and performed before administration of the study drug if it is the day of study drug administration. Each score will be recorded in the (e)CRF.

## 9.1.11 Laboratory Test

Clinical laboratory test items as shown in Table 9.b will be determined. The test samples will be collected before administration of the study drug if it is the day of study drug administration. All samples will be handled in accordance with the separately specified procedures. The maximum amount of blood sampling will be approximately 19 mL at each visit.

Table 9.b Laboratory tests

| Blood biochemistry | | |
|---|---|---|
| Albumin Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Alkaline phosphatase (ALP) Amylase Glucose Note1) Total bilirubin Total protein g-glutamyl transpeptidase (γ-GTP) | | Total cholesterol Triglyceride 1) Creatinine Blood urea nitrogen (BUN) Uric acid Potassium Sodium Calcium Phosphorus Magnesium Chloride |
| Hematology | | Urinalysis |
| Red blood cells White blood cells Hemoglobin Hematocrit Platelets | Neutrophils Eosinophils Basophils Lymphocytes Monocytes | Qualitative (glucose, protein, occult blood, bilirubin, ketone body) Urine pH Urine specific gravity |
| Serum immunological test (only at screening) 2) | | Urine pregnancy test (only in female subjects of childbearing potential) |
| HBs antigen/antibody, HBc antibody, HCV antibody<br>HIV antibody | | Human chorionic gonadotrophin (hCG) |
| Inflammatory markers | S | |
| C-reactive protein (CRP | 2) | |

- 1) The samples should be preferably collected under fasted conditions.
- 2) The test results of the serum immunological tests should be reported to subjects directly by investigator, and not be provided to the sponsor.

The above laboratory test items will be determined at the laboratory site for the study except urine pregnancy tests. The urine pregnancy tests will be performed at the study sites. Investigator will assess and retain the clinical laboratory test results reported.

If subjects experience ALT or AST >3×ULN, follow-up laboratory tests (at a minimum, ALP, ALT, AST, total bilirubin,  $\gamma$ -GTP, and INR) should be performed preferably within 48 to 72 hours or within 7 days at the latest after the blood sampling (see Section 7.5 and Section 10.2.3).

If the ALT or AST remains elevated >3×ULN on these 2 consecutive occasions, the investigator must contact the Medical Monitor for consideration of additional testing, close monitoring, possible discontinuation of the study drug, discussion of the relevant subject details and possible alternative etiologies.

Investigators will retain references of the clinical laboratory tests and their tracking.

#### 9.1.12 Contraception and Pregnancy Avoidance Procedure

During the period from the time of signing on the informed consent form to 6 months after the last dose of the study drug, female subjects of childbearing potential (who have no history of sterilization or have menstruation within previous 2 years) must use proper contraception. In addition, during the period from the time of signing on the informed consent form to 6 month after the last dose of the study drug, male subjects without history of sterilization and whose female partner has child bearing potential must prevent pregnancy. Such subjects will be provided with information on acceptable methods of contraception as part of the subject informed consent process, and will be asked to sign a consent form stating that they understand the requirements for avoidance of pregnancy during the course of the study. During the course of the study, the specified urine pregnancy tests will be performed, and subjects will receive continued guidance with respect to avoiding pregnancy.

Urine pregnancy tests performed at screening and at immediately before the first dose of the study drug should be confirmed to show negative.

In addition, male subject must be advised not to donate sperm from the time of signing on the informed consent form to 6 months after the last dose of the study drug.

## 9.1.13 Pregnancy

If any subject is found to be pregnant during the study, she should be withdrawn and any sponsor-supplied study drugs should be immediately discontinued.

Any pregnancies occurred during the period from the first dose of the study drug (Visit 2) to 6 months after the last dose of the study drug should be reported, using the given report form, to the contact listed in the Annex. In addition, any pregnancies in the partner of a male subject during the period from the first dose of the study drug (Visit 2) to 6 months after the last dose of the study drug should also be recorded following authorization from the subject's partner.

Should the pregnancy occur during or after administration of the blinded drug, the investigator must inform the subject of their right to receive treatment information. Upon subject's request, the investigator will open the Emergency Key. Subjects revealed not to have received MLN0002 in the study are not required to be followed.

Upon consent with the female subject or the female partner of the male subject, the investigator should inform their physician (an obstetrician) that the subject/female partner of the subject was participating in the clinical study at the time of conception with details of treatment the subject received (blinded or unblinded, as applicable).

All reported pregnancies will be followed up to final outcome, using the pregnancy form. The outcome, including any premature termination, must be reported to the sponsor. An evaluation after the birth of the child will also be conducted.

#### 9.1.14 ECG Procedure

A standard 12-lead ECG will be recorded. The investigator (or a qualified observer at the study site) will interpret the ECG using 1 of the following categories: within normal limits, abnormal but not clinically significant, or abnormal and clinically significant.

#### 9.1.15 PML Evaluation

PML will be evaluated based on the PML checklists (Appendix D), which will be performed before administration of the study drug if it is the day of study drug administration.

At first, the subjective symptoms will be checked by use of the Subjective PML checklist. When any subjective symptoms are recognized, the corresponding objective findings will be checked by use of the Objective PML checklist. When any abnormalities are found in the objective findings as well, the subject will be evaluated in accordance with the algorithm for subject evaluation in the PML checklists.

The evaluation result based on the PML checklists will be recorded in the (e)CRF. Any subjective symptoms or objective findings found in the PML checklists will be collected as AEs as well.

#### 9.1.16 Tuberculosis test

As a sample for tuberculosis test, 7 mL of the whole blood will be collected. The laboratory site for the study will collect the sample to conduct tuberculosis test by means of T-SPOT. The tuberculosis test using QuantiFERON may be conducted, when routinely employed in the study site. The test results, i.e. positive, negative, indeterminate or indeterminable, will be recorded in the (e)CRF.

#### 9.1.17 Chest Imaging Procedure

Existence of findings of tuberculosis will be confirmed by the chest X-ray or chest CT. The imaging performed within 3 months before evaluation as a part of general practice not as a test for the study may be used, if available. Date of Examination and existence of findings of tuberculosis will be recorded in the (e)CRF.

Of note, the imaging obtained before acquisition of the informed consent may be used at screening.

#### 9.1.18 Pharmacogenomic Sample Collection

For exploratory research to identify a predictable marker of drug response, 5 mL of the whole blood will be once collected as a pharmacogenomic sample from subjects entered into the induction phase and who agreed with the pharmacogenomic research at the earliest possible time during the period from Visit 2 to the end of the study.

However, the pharmacogenomic samples will not be collected from subjects with a history of an allogeneic bone marrow transplantation.

See the separately specified written procedure for collecting, handling, and storing the pharmacogenomic samples.


## 9.1.19 Pharmacokinetic Sample Collection and Analysis

Pharmacokinetic samples will be collected only in study sites with a cooled centrifuge. In these study sites, 3 mL of the venous blood will be collected for determination of serum MLN0002 concentration. At the visit for study drug administration, the blood should be sampled immediately before administration, where possible. The date and time of the blood sampling will be recorded in the (e)CRF.

The collected blood will be left standing at room temperature for approximately 30 minutes and centrifuged at 3,000 rpm at 4°C for 10 minutes. The obtained serum will be cryopreserved in a preset freezer at a temperature of  $\leq$ -20°C until collection. The samples will be handled in accordance with the separately specified procedures.

Serum MLN0002 concentration will be determined in PPD by means of Enzyme-Linked ImmunoSorbent Assay (ELISA). However, samples of subject who have not received MLN0002 throughout the induction and maintenance phases will not be determined.

## 9.1.20 Sample Collection for the HAHA/Neutralizing Antibody Test

Samples for the HAHA/neutralizing antibody test will be collected only in study sites with a cooled centrifuge. In these study sites, 5 mL of the venous blood will be collected for the HAHA/neutralizing antibody test. At the visit for study drug administration, the blood should be sampled immediately before administration, where possible. The date and time of the blood sampling will be recorded in the (e)CRF.

The collected blood will be left standing at room temperature for approximately 30 minutes and centrifuged at 3,000 rpm at 4°C for 10 minutes. The obtained serum will be cryopreserved in a preset freezer at a temperature of  $\leq$ -20°C until collection. The samples will be handled in accordance with the separately specified procedures.

Serum concentration of HAHA will be determined in PPD by means of ELISA. However, samples of subjects who have not received MLN0002 throughout the study will not be determined.

Furthermore, the serum neutralizing antibody will be determined only for the HAHA-positive samples. The serum neutralizing antibody will be determined in PPD by means of the Cell Based Assay.

## 9.1.21 Record of Subjects Who Withdrew during the Screening Phase

The (e)CRFs will be documented for all subjects who signed the informed consent and withdrew during the screening phase. The primary reason for screen failure is recorded in the (e)CRF by the following categories:

- Pretreatment Event/AE
- Did not meet inclusion criteria or met exclusion criteria <specify the reason>
- Major protocol deviation

- Lost to follow-up
- Voluntary withdrawal <specify the reason>
- Study termination
- Pregnancy
- Other <specify the reason>

The Subject Identification Codes applied to subjects who withdrew during the screening phase will not be reused.

#### 9.1.22 Enrollment into the induction Phase

Only subjects who meet all of the inclusion criteria and none of the exclusion criteria are eligible for enrollment into the induction phase at Week 0 (Visit 2). At enrollment into the induction phase, the following information will be registered on the website of the registration center where the study drug number to be dosed at Week 0 (Visit 2) will be provided.

- Treatment history with anti-TNFα antibodies
- Concomitant use of immunomodulators (AZA, 6-MP or MTX)
- Concomitant use of corticosteroids
- The subject diary data for calculation of the CDAI score at Week 0 (Visit 2)

# 9.1.23 Registration of the Results of the Primary Efficacy Endpoint in the Induction Phase/Enrollment into the Maintenance Phase

The subject diary data for calculation of the CDAI score at Week 10 (Visit 5) will be registered on the website of the registration center, by which adjudication results for clinical response/no-response may be obtained. Only CDAI-70 responders at Week 10 will be enrolled into the maintenance phase at Week 14 (Visit 6). At enrollment into the maintenance phase, the study drug number to be dosed at Week 14 (Visit 6) will be obtained on to the website of the registration center.

See Section 9.1.24 for non-responders at Week 10.

#### 9.1.24 Enrollment into the Open-label Cohort

Non-responders at Week 10 may be enrolled into the open-label cohort at Week 10 (Visit 5). In addition, either subjects who experienced disease worsening or received rescue treatments during the maintenance phase, or completed Week 60 of the maintenance phase may be enrolled into the open-label cohort. However, subjects who withdrew before the examination at Week 10 (Visit 5), or subjects who respond at Week 10 and withdrew before enrollment into the maintenance phase at Week 14 (Visit 6) are not allowed to be enrolled into the open-label cohort.

The procedures for enrollment into the open-label cohort is provided below;

- Non-responders at Week 10:
  - Non-responders at Week 10 will be judged whether to be enrolled into the open-label cohort after completion of examination at Week 10 (Visit 5). For enrolled into the open-label cohort, the study drug number to be dosed at Week 0x (Visit 1x) will be obtained on the website of the registration center.
- Subject experienced disease worsening or received rescue treatments during the maintenance phase:
  - Subjects who experienced disease worsening or received rescue treatments during the maintenance phase will be judged whether to be enrolled into open-label phase after completion of the evaluation at withdrawal of the maintenance phase. However, these subjects will be enrolled into open-label phase 3 to 9 weeks after the last dose in the maintenance phase. For enrollment into the open-label cohort, the study drug number to be dosed at Week 0x (Visit 1x) will be obtained on the website of the registration center.
- Subjects completed Week 60: Subjects who completed Week 60 will be judged whether to be enrolled into the open-label cohort after completion of examination at Week 60 (Visit 18). For enrollment into the open-label cohort, the study drug number to be dosed at Week 0x (Visit 1x) will be obtained on the website of the registration center.

## 9.2 Study Drug Compliance

The study drugs dosed to the subjects will be recorded in the (e)CRF for the dates, times of start/end of the infusion. When infusion of a study drug was not completed, dosage and reasons for dose incomplete will be recorded in the (e)CRF.

#### 9.3 Schedule of Observations and Procedures

The schedule for all study-related procedures for all evaluations is shown in Appendix A. Assessments should be completed at the designated visit/time point(s).

## 9.3.1 The Screening Phase (Visit 1)

Physical examination and tests are conducted 21 to 7 days before the first dose of the study drug. Subjects will be screened in accordance with predefined inclusion and exclusion criteria as described in Section 7.0. See Section 9.1.21 for procedures for documenting screening failures.

Procedures to be completed at Screening Phase (Visit 1) include:

- Informed consent
- Demographic data, body height, medical history, pretreatment drugs, and complications
- Physical examination, vital signs
- Body weight

- ECG
- Chest Imaging Procedure\*
- Tuberculosis test
- PML checklists
- Laboratory tests (see Appendix A for test items)
- Concomitant drugs and treatments
- PTEs assessment
  - \* Not required when a chest image performed within 3 months is available (the image taken outside the study and/or prior to the informed consent date is acceptable).

#### 9.3.2 Induction Phase

## 9.3.2.1 Baseline Evaluation/Enrollment into the induction Phase (Visit 2)

Subjects will be screened in accordance with predefined inclusion and exclusion criteria as described in Section 7.0. Subjects who meet all of the inclusion criteria and none of the exclusion criteria are eligible for enrollment into the induction phase at Week 0 (Visit 2) as per Section 9.1.22. See Section 9.1.21 for procedures for documenting subjects not eligible for enrollment into the induction phase.

Tests/observations/assessments to be performed at Week 0 (Visit 2) include:

- Physical examination, vital signs
- Body weight
- ECG
- PML checklists
- Laboratory tests (see Appendix A for test items)
- CDAI score (including determination of Ht level. See Section 9.1.9 for details)
- Check of the patient diary
- IBDO
- Blood sampling for HAHA /neutralizing antibody test
- Blood sampling for pharmacogenomics (in subjects providing agreements)
- Concomitant drugs and treatments
- Evaluation of Pretreatment Event/AE
- Issuance of study drug numbers/administration


## 9.3.2.2 Administration in the Induction Phase (Visits 3 and 4)

Procedures to be completed at Week 2 (Visit 3) and Week 6 (Visit 4) include:

- Physical examination, vital signs
- Body weight
- PML checklists
- Laboratory tests (see Appendix A for test items)
- CDAI score (including determination of Ht level. See Section 9.1.9 for details)
- Check of the patient diary
- Blood sampling for serum drug concentration
- Concomitant drugs and treatments
- Evaluation of AEs
- Issuance of study drug numbers/administration

## 9.3.2.3 Evaluation of Primary Efficacy Endpoint (Visit 5)/Withdrawal during the Induction Phase

Procedures to be completed at Week 10 (Visit 5) include: The same procedures will be completed at the earliest possible visit for subjects who withdrew in the course of the induction phase.

- Physical examination, vital signs
- Body weight
- ECG
- Laboratory tests (see Appendix A for test items)
- CDAI score (including determination of Ht level. See Section 9.1.9 for details)
- Check of the patient diary
- IBDQ
- Blood sampling for HAHA /neutralizing antibody test
- Blood sampling for serum drug concentration
- Concomitant drugs and treatments
- Evaluation of AEs

An adjudication result for clinical response/not-response at Week 10 (Visit 5) will be obtained from the registration center. Responders will be enrolled into the maintenance phase at Week 14 (Visit 6). Non-responders may be enrolled into the open-label cohort at Week 10 (Visit 5).

#### 9.3.3 Maintenance Phase

## 9.3.3.1 Enrollment into the maintenance Phase (Visit 6)

Responders at Week 10 (Visit 5) will be enrolled into the maintenance phase at Week 14 (Visit 6) in accordance with Section 9.1.23.

Procedures to be completed at Week 14 (Visit 6) include:

- Physical examination, vital signs
- Body weight
- PML checklists
- Laboratory tests (see Appendix A for test items)
- CDAI score (including determination of Ht level. See Section 9.1.9 for details)
- Check of the patient diary
- IBDO
- Blood sampling for serum drug concentration
- Concomitant drugs and treatments
- Evaluation of AEs
- Issuance of study drug numbers/administration

## 9.3.3.2 Administration in the Maintenance Phase (Visits 7 through 17)

Procedures to be completed at Week 18 (Visit 7) through Week 58 (Visit 17) include:

- Physical examination, vital signs
- Body weight
- PML checklists (only at Visits 8, 10, 12, 14 and 16)
- Laboratory tests (only at Visits 8, 10, 12, 14 and 16. See Appendix A for test items)
- CDAI score (including determination of Ht level. See Section 9.1.9 for details)
- Check of the patient diary
- IBDQ (only at Visit 12)
- Blood sampling for HAHA/neutralizing antibody test (only at Visit 10)
- Blood sampling for serum drug concentration (only at Visits 8 and 10)
- Concomitant drugs and treatments

- Evaluation of AEs
- Issuance of study drug numbers/administration (only at Visits 8, 10, 12, 14 and 16)

# 9.3.3.3 Evaluation of Primary Efficacy Endpoint in the Maintenance Phase (Visit 18)/Withdrawal during the Maintenance Phase

Procedures to be completed at Week 60 (Visit 18) include: The same procedures will be completed at earliest possible visit for subjects who withdrew in the course of the maintenance phase.

- Physical examination, vital signs
- Body weight
- ECG
- Laboratory tests (see Appendix A for test items)
- CDAI score (including determination of Ht level. See Section 9.1.9 for details)
- Check of the patient diary
- IBDO
- Blood sampling for HAHA /neutralizing antibody test
- Blood sampling for serum drug concentration
- Concomitant drugs and treatments
- Evaluation of AEs

Subjects who completed the examination at Week 60 (Visit 18) may be enrolled into the open-label cohort at Week 60 (Visit 18). Furthermore, subjects who experienced disease worsening or received rescue treatments during the maintenance phase may be enrolled into the open-label cohort after completion of the evaluation at withdrawal of the maintenance phase.

#### 9.3.4 Open-label Cohort

## 9.3.4.1 Enrollment into the open-label cohort (Visit 1x)

Subjects who have been decided to be enrolled into the open-label cohort as per Section 9.1.24 will be enrolled into the open-label cohort. Procedures to be completed at Week 0x (Visit 1x) include:

- PML checklists
- Concomitant drugs and treatments
- Evaluation of AEs
- Issuance of study drug numbers/administration

## 9.3.4.2 Administration in the Open-label Cohort (Visits 2x through 24x)

Procedures to be completed at Week 2x (Visit 2x) through Week 90x (Visit 24x) include:

- Physical examination, vital signs
- Body weight
- PML checklists (only at Visits 2x, 3x, 5x, 7x, 9x, 11x, 13x, 15x, 17x, 19x, 21x and 23x)
- Laboratory tests (only at Visits 2x, 3x, 5x, 7x, 9x, 11x, 13x, 15x, 17x, 19x, 21x and 23x. See Appendix A for test items)
- CDAI score (including determination of Ht level. See Section 9.1.9 for details)
- Check of the patient diary
- Blood sampling for HAHA /neutralizing antibody test (only at Visits 4x, 9x and 17x)
- Concomitant drugs and treatments
- Evaluation of AEs
- Issuance of study drug numbers/administration (only at Visits 2x, 3x, 5x, 7x, 9x, 11x, 13x, 15x, 17x, 19x, 21x and 23x).

# 9.3.4.3 The Final Evaluation of the Open-label Cohort (VIST 25x)/Withdrawal during the Open-label Cohort

Procedures to be completed at Week 94x (Visit 25x) include: The same procedures will be completed at the earliest possible visit for subjects who withdrew in the course of the open-label cohort.

- Physical examination, vital signs
- Body weight
- ECG
- PML checklists
- Laboratory tests (see Appendix A for test items)
- CDAI score (including determination of Ht level. See Section 9.1.9 for details)
- Check of the patient diary
- Blood sampling for HAHA /neutralizing antibody test
- Concomitant drugs and treatments
- Evaluation of AEs

• Issuance of study drug numbers/administration (not for subjects who withdrew from the open-label cohort)

#### 9.3.5 The Unscheduled Visits

The following procedures will be preferably completed at the unscheduled visits of any subjects who received the study drug due to worsening of CD, etc., if any.

- Body weight
- CDAI score (including determination of Ht level. See Section 9.1.9 for details)
- Check of the patient diary
- Concomitant drugs and treatments
- Evaluation of AEs

Besides the above, additional tests may be performed as needed.

The subject's applicability to the disease worsening criteria (see Section 3.1 for definition) will be judged in consideration of test results performed at the unscheduled visit as well. In such cases, the interval between visits will be not less than 1 week, where possible.

## 9.3.6 Predefined Study Completion

The same examination as those to be performed at Week 94x (Visit 25x) will be performed at study completion predefined at 46 weeks after the last subject enrollment into the open-label cohort.

The sponsor will inform the investigator of the scheduled study completion date well before the date.

Upon receipt of notice of the scheduled study completion date, the investigator will decide the termination visits for each subjects to undergo the same evaluation as those scheduled at Week 94x (Visit 25x).

#### 9.3.7 At 16 weeks after the Last Dose

The following evaluation will be conducted at 16 weeks after the last dose of the study drug for all subjects who received the study drug. Even when the study will be terminated before 16 weeks have passed after the last dose of the study drug, the same evaluation will also be conducted in principle.

For all subjects who received the study drug, the investigator must complete the End of Study (e)CRF page.

- Physical examination, vital signs
- Body weight

- ECG
- Chest Imaging Procedure\*
- PML checklists
- Laboratory tests (see Appendix A for test items)
- Blood sampling for HAHA /neutralizing antibody test
- Concomitant drugs and treatments
- Evaluation of AEs
  - \* Not required when a chest image performed within 3 months is available (the image taken outside the study is acceptable).

## 9.3.8 Post Study Care

The study drugs will not be provided after the last dose.

## 9.4 Retention and Disposal of Biological Samples

The samples of 5 mL of the whole blood collected for Pharmacogenomic Research will be cryopreserved in PPD (Annex 1).

The retention period should be 20 years from the first sampling day for Pharmacogenomic Research in the study.

Upon subject's request of disposal of his/her samples during the retention period, the study site will request PPD to dispose of the samples via the sponsor as per the procedures. PPD will dispose of the samples in accordance with the procedures, which will be reported to the study site and the sponsor. However, the above is not applicable, when all documents (e.g., medical records) to be used for identification of subjects have been disposed of after study termination, so that any samples and subjects are impossible to be linked together.

Of note, even though the above linkage may be possible, when Pharmacogenomic Research has been conducted already, the sponsor may keep the anonymized results of the Pharmacogenomic Research with the residual samples disposed.

The sponsor will create a necessary written procedure as establishing a necessary control system for protecting subjects' personal information and predefining the standards for collection, retention and disposal of samples.

#### 9.5 Follow-Up Survey

In the study, the follow-up survey will be conducted via telephone, etc., by using the follow-up survey form (Appendix E) every 6 months up to 2 years (maximum) after the last dose of the study drug or until the marketing approval date of the drug, whichever comes earlier, for any subjects

who received the study drug (including subjects who withdrew). The follow-up survey include the following items. Of note, the follow-up survey forms will be collected by the sponsor.

The survey to be completed at 6, 12, 18 and 24 months<sup>4</sup> after the last dose of the study drug:

- Diagnoses of colon dysplasia, cancer, lymphoma or other types of cancer
- Diagnoses of PML
- Enterectomy

The survey to be completed only once at 6 months<sup>4</sup> after the last dose of the study drug:

- Diagnoses of infection requiring hospitalization
- Female subjects: pregnancy
- Male subjects: pregnancy of his female partner

\_

<sup>&</sup>lt;sup>4</sup>The window is  $\pm 1$  month.

#### 10.0 PRETREATMENT EVENTS AND ADVERSE EVENTS

#### 10.1 Definitions

#### 10.1.1 PTEs

A PTE is defined as any untoward medical occurrence in a subject who has signed the informed consent to participate in a study but prior to administration of any study drug; it does not necessarily have to have a causal relationship with study participation.

#### 10.1.2 AEs

An AE is defined as any untoward medical occurrence in a study subject who received a drug (including a study drug); it does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug.

#### 10.1.3 Additional Points to Consider for PTEs and AEs

An untoward finding generally may include:

- A new diagnosis or those representing unexpected worsening of a pre-existing condition (intermittent events of pre-existing conditions of an underlying disease should not be considered PTEs or AEs.)
  - Intermittent events of pre-existing conditions of an underlying disease in the study include some CD-specific symptoms such as diarrhea or abdominal pain. These symptoms, which may be sustained or varied in the course of the study depending on medical histories of each subject, will be considered as medically-predictable clinical symptoms in the disease addressed in the study, and therefore, not be subjected for collection of AEs. These symptoms corresponding to disease activity will be assessed as a part of the CDAI score. However, worsening of disease activity (e.g., abdominal pain aggravated beyond a normal range, or newly-observed symptoms or findings) will be collected as AEs. Onset or worsening of extra-intestinal manifestations in the course of the study will be collected as AEs.
- Those requiring therapeutic intervention
- Those requiring an invasive diagnostic procedure
- Those requiring discontinuation or dose modification of the study drug or a concomitant drug
- Those considered as unfavorable by the investigator for any reason.

Diagnoses vs signs and symptoms:

PTEs and AEs (hereinafter called as PTEs/AEs) will be described as diagnoses. Accompanying signs (including abnormal laboratory values or ECG findings) or symptoms should NOT be

recorded as PTEs/AEs. If a diagnosis is unknown, sign(s) or symptom(s) should be recorded appropriately as PTEs/AEs.

#### Laboratory values and ECG parameters:

Changes in laboratory values or ECG parameters are considered as PTEs/AEs only when they are judged to be clinically significant (i.e., when some action or intervention is required or if investigator judges the change as being beyond the range of normal physiologic fluctuation). A laboratory re-test and/or continued monitoring of an abnormal value are not considered an intervention. In addition, repeated or additional noninvasive testing for verification, evaluation or monitoring of an abnormality is not considered an intervention.

If abnormal laboratory values or ECG findings are the result of pathology for which there is an overall diagnosis (e.g., increased creatinine in renal failure), the diagnosis only should be reported appropriately as a PTE or as an AE.

## Pre-existing conditions:

Any pre-existing diseases or conditions prior to acquisition of the informed consent will be recorded as complications not as PTEs/AEs. Baseline evaluations (e.g., laboratory tests, ECG, X-rays etc.) should NOT be recorded as PTEs unless related to study procedures. However, abnormal findings caused by the baseline evaluation (e.g., internal hemorrhage at blood sampling) are recorded as PTEs to be entered in the (e)CRF. Investigators should ensure that the event term recorded captures the change in the condition (e.g., "worsening of...").

If a subject has a pre-existing episodic condition (e.g., asthma, epilepsy), any occurrence of an episode should be captured as a PTE/AE only when the episodes become more frequent, serious or severe in nature, that is, investigators should ensure that the AE term recorded captures the change in the condition from Baseline (e.g., "worsening of..."). If a subject has a degenerative concurrent condition (e.g., cataracts, rheumatoid arthritis), worsening of the condition should be captured as a PTE/AE only when occurring to a greater extent to that which would be expected. Again, investigators should ensure that the AE term recorded captures the change in the condition (e.g., "worsening of...").

#### Worsening of PTEs/AEs:

If the subject experiences a worsening or complication of a PTE after starting administration of the study drug, the worsening or complication should be recorded appropriately as an AE. Investigators should ensure that the AE term recorded captures the change in the condition (e.g., "worsening of...").

If the subject experiences a worsening or complication of an AE after any change in the study drug, the worsening or complication should be recorded as a new AE. Investigators should ensure that the AE term recorded captures the change in the condition (e.g., "worsening of...").

#### Changes in severity of AEs/Serious PTEs:

If the subject experiences changes in severity of an AE/serious PTE, the event should be captured once with the maximum severity recorded.

## Preplanned surgeries or procedures:

Preplanned procedures (surgeries or therapies) that were scheduled prior to the time of signing on the informed consent form are not considered PTEs/AEs. However, if a preplanned procedure is performed early (e.g., as an emergency) due to a worsening of the pre-existing condition, the worsening of the condition should be captured appropriately as a PTE/AE. Complications resulting from any planned surgery should be reported as AEs.

#### Elective surgeries or procedures:

Elective procedures performed where there is no change in the subject's medical condition should not be recorded as PTEs/AEs, but should be documented in the subject's source documents. Complications resulting from an elective surgery should be reported as AEs.

## Insufficient clinical response (lack of efficacy):

Insufficient clinical response, efficacy, or pharmacologic action should NOT be recorded as an AE. Investigator must make the distinction between exacerbation of pre-existing illness and lack of therapeutic efficacy.

#### Overdose:

Cases of overdose with any drug are NOT considered AEs, but instead will be documented on an Overdose page of the (e)CRF. Any manifested side effects at overdose will be considered AEs and will be recorded on the AE page of the (e)CRF.

#### 10.1.4 **SAEs**

SAEs are defined as the following out of any untoward medical occurrence in a study subject who received a drug (regardless of dosages);

- 1. Results in DEATH.
- 2. Is LIFE THREATENING\*
- 3. Requires inpatient HOSPITALIZATION or prolongation of existing hospitalization.
- 4. Results in persistent or significant DISABILITY/INCAPACITY.
- 5. Leads to a CONGENITAL ANOMALY/BIRTH DEFECT.
- 6. Other medically significant conditions
  May require intervention to prevent the above items 1 through 5, or may expose the subject to
  danger, even though the event is not immediately life-threatening or fatal or does not result in
  hospitalization. That includes any events or synonyms described in the Takeda Medically
  Significant AE List (Table 10.a).

\*The "life-threatening" here represents that life of the subject was threatened by onset of the event, and does not represent hypothetically that a more sever event might cause death.

## Table 10.a Takeda Medically Significant AE List

| Acute respiratory failure / acute respiratory distress syndrome | Hepatic necrosis Acute liver failure |
|---|---|
| Torsade de pointes / ventricular fibrillation / | Anaphylactic shock |
| ventricular tachycardia | Acute renal failure |
| Malignant hypertension | Pulmonary hypertension |
| Convulsive seizures | Pulmonary fibrosis |
| Agranulocytosis Aplastic anemia | Neuroleptic malignant syndrome / malignant hyperthermia |
| Toxic epidermal necrolysis/Stevens-Johnson | Spontaneous abortion / stillbirth and fetal death |
| syndrome | Confirmed or suspected transmission of infectious agent by a medicinal product |
| | Confirmed or suspected endotoxin shock |

PTEs that fulfill 1 or more of the serious criteria above are also to be considered SAEs and should be reported and followed up in the same manner (see Sections 10.2.2 and 10.2.3).

## 10.1.5 Intensity of PTEs and AEs

Intensity of PTEs/AEs will be classified/defined as per the following.

| Mild: | The event is transient and easily tolerated by the subject. |
|---|---|
| Moderate: | The event causes the subject discomfort and interrupts the subject's usual activities. |
| Severe: | The event causes considerable interference with the subject's usual activities. |

#### 10.1.6 Causality of AEs

Causal relationship between AEs and study drugs will be classified/defined as per the following.

| Related: | An AE that follows a temporal sequence from administration of a drug (including the course after withdrawal of the drug), or for which possible involvement of the drug can be argued, although factors other than the drug, such as underlying diseases, complications, concomitant drugs, and concurrent treatments, may also be responsible. |
|---|---|
| Not Related: | An AE that does not follow a temporal sequence from administration of a drug and/or that can reasonably be explained by other factors, such as underlying diseases, complications, concomitant drugs, and concurrent treatments. |

## **10.1.7** Relationship to Study Procedures

Relationship (causality) to study procedures should be determined for all PTEs/AEs. The relationship should be assessed as Yes if the investigator considers that there is reasonable possibility that an event is due to a study procedure. Otherwise, the relationship should be assessed as Not Related.

#### 10.1.8 Start Dates

Onset dates of PTEs/AEs will be decided as per the following criteria;

| PTEs/AEs | Onset Dates |
|---|---|
| Signs, symptoms or disease (diagnoses) | The date when the subject or the investigator was firstly aware of the sign/symptom. |
| Asymptomatic disease | The date of the definitive diagnosis on or after the diagnostic examination, even when any obsolete findings or other estimated onset time was found in the examination. |
| Worsening of complications or PTEs | The date when the subject or the investigator was firstly aware of the worsening of the disease or symptoms. |
| Newly-indicated abnormal laboratory values in values shown to be normal in the baseline test after acquisition of the informed consent (PTEs) Newly-indicated abnormal laboratory values after the first dose of the study drug (AEs) | The date of the examination in which the clinically relevant abnormality was found. |
| Worsening of abnormal laboratory values found in the baseline test after acquisition of the informed consent (PTEs) Worsening of abnormal laboratory values found at the first dose of the study drug (AEs) | The date of the examination in which the medically-judged obvious increase/decrease/elevation/reduction was found by change of the test results. |

#### **10.1.9 Stop Date**

The stop date is defined as the date when the PTE/AE was recovered/resolved (including recovered/resolved with sequelae), or the date of death when caused by the PTE/AE. PTEs/AEs, which may not be confirmed for recovery/resolution at the study termination, will be judged as ongoing.

#### **10.1.10** Frequency

Episodic AEs/serious PTE (e.g., vomiting) or those which occur repeatedly over a period of consecutive days are "intermittent." All other events will be recorded as "ongoing."

## 10.1.11 Action Concerning Study Drug

Action concerning study drug will be classified/defined as per the following.

| Drug withdrawn | A study drug is stopped due to the particular AE. |
|---|---|
| Dose not changed | When the dose was not changed after the AE, when the dose discontinuation/reduction/increase was due to other AEs than the AE, or when the dose suspension/reduction/etc., was due to other reason (e.g., carelessness of the subject) than AEs. |
| Unknown | Only to be used if it has not been possible to determine what action has been taken. |

| A study drug was stopped for a reason other than the particular AE eg, the study has been terminated, the subject died, dosing with study drug was already stopped before the onset of the AE. |
|---|
|---|

#### **10.1.12** Outcome

Outcome of PTEs/AEs will be classified/defined as per the following.

| Classification | Criteria for judgment |
|---|---|
| Recovered/Resolved | Recovery or resolution of the symptom/finding |
| | <ul> <li>Recovery to the normal value, the value before the first dose (for AEs), or the value at<br/>baseline after acquisition of the informed consent (for PTEs).</li> </ul> |
| Recovering/Resolving | The severity is lowered by one or more degree(s) |
| | <ul> <li>The diagnosis or signs/symptoms has almost disappeared</li> </ul> |
| | <ul> <li>The abnormal laboratory value improved, but has not returned to the normal range or<br/>to baseline.</li> </ul> |
| | <ul> <li>The subject died from a cause other than the particular AE/serious PTE with the<br/>condition remaining "recovering/resolving."</li> </ul> |
| Not recovered/<br>not resolved | - There is no change in the diagnosis, signs or symptoms; |
| | <ul> <li>The intensity of the diagnosis, signs/ symptoms or laboratory value on the last day of<br/>the observed study period has got worse than when it started;</li> </ul> |
| | - Irreversible congenital anomaly |
| | <ul> <li>The subject died from another cause with the particular AE/serious PTE state<br/>remaining "Not recovered/not resolved."</li> </ul> |
| Resolved with sequelae | Resulting in dysfunction obstructing daily activity |
| Fatal | The PTE/AE are considered to have a direct relationship with the death. |
| | <ul> <li>The "direct relationship" here represents that the PTE/AE was the cause of the death,<br/>or clearly contributed to the death.</li> </ul> |
| | <ul> <li>Outcome should not be recorded as death for the PTE/AE not adjudicated<br/>(judged/estimated) as the direct cause of death in the same subject.</li> </ul> |
| | <ul> <li>The date of death will be recorded for fatal outcomes.</li> </ul> |
| Unknown | <ul> <li>The course of the AE/serious PTE cannot be followed up due to hospital change or<br/>residence change at the end of the subject's participation in the study.</li> </ul> |

#### 10.2 Procedures

## 10.2.1 Collection and Reporting of AEs

#### 10.2.1.1 PTE and AE Collection Period

PTEs will be continuously collected during the period from acquisition of the informed consent to the first dose of the study drug (Visit 2), or until withdrawal when decided before the first dose of the study drug.

AEs will be continuously collected during the period from the first dose of the study drug (Visit 2) to the end-of-study examination at 16 weeks after the last dose of the study drug.

#### 10.2.1.2 PTE and AE Reporting

Subjects may report PTEs/AEs occurring at any other time during the study. PTEs/AEs not emerging at visit will be obtained from subjects with questions such as "How was your condition after the last visit?."

Investigators will follow all subjects who developed a serious PTE until recovery/resolution of the event or recovery of the clinically relevant abnormal test value to the baseline value after acquisition of the informed consent, or otherwise (for persistent/irreversible PTEs) until establishment of sufficient rationale for the observed change. Subjects who developed not-serious PTEs are not required to be followed irrespective of relationship with study procedures in the protocol.

Investigators will follow all subjects who developed an AE (with or without relationship with the study drug) until recovery/resolution of the event or recovery of the clinically relevant abnormal test value to the value before the first dose of the study drug, or otherwise (for persistent/irreversible AEs) until establishment of sufficient rationale for the observed change. All PTEs/AEs should be recorded in the (e)CRF. For a PTE/AE, the name, onset date, recovery/resolution date, start period, frequency, severity, causal relationship with the study drug (related/not-related), disposition of the study drug, outcome, causal relationship with the study procedures (if related, the possible causal procedure), and seriousness will be recorded.

For AEs that occurred during infusion of the study drug or the period from initiation to 1 hour after completion of infusion, onset time and association with infusion will be recorded in the (e)CRF.

AEs/serious PTEs will be followed until the PTE/AE is recovered/resolved or the investigator judges not to follow them any longer.

## 10.2.2 Collection and Reporting of SAEs

When a SAE occurs during the AE collection period, it should be reported according to the following procedure: PTEs that fulfill 1 or more of the serious criteria described in Section 10.1.4 are also considered as SAEs to be reported and followed in the same manner.

Investigators should report the SAE within 1 working day after onset of the SAE or receipt of the notice of the event onset from a subject, etc., to the sponsor (see the Annex for contacts). Additionally, the investigator should submit the detailed formal reports within 10 calendar days.

Of note, the following is specified as the essential items to be reported within 1 working day, however, other items should be provided as much as possible.

- A short description of the event and the reason why the event is categorized as serious.
- Subject Identification Code
- Investigator's name.

- Name of the study drugs
- Causality assessment

Any SAE spontaneously reported to the investigator following the AE collection period (including the follow-up survey period) should be reported to the sponsor.

## 10.2.3 Drug-induced Liver Function Test Abnormal Possibly Leading to Sever Liver Disorder

If a subject is noted to have ALT or AST >3 ×ULN and total bilirubin >2 ×ULN for which an alternative etiology has not been identified, the event should be recorded as an SAE and reported as per Section 10.2.2. The investigator must contact the Medical Monitor for discussion of the relevant subject details and possible alternative etiologies, such as acute viral hepatitis A or B or other acute liver disease. Follow-up laboratory tests as described in Section 9.1.11 must also be performed. These abnormal liver function test values, when judged not to be explained by any other factors, should be reported as SAEs (see Section 10.2.2).

#### 10.3 Follow-up of SAEs

For information obtained after submission of the detailed report, the investigator should describe them in a copy of the submitted SAE Report Form or as an independent document in order to be submitted to the contact listed in the Annex. Copies of any relevant data from the hospital notes (e.g., ECGs, laboratory tests, discharge summary, postmortem results) should be sent to the addressee, if requested.

All SAEs should be followed up until resolution or permanent outcome of the event.

#### 10.3.1 SAE Reports to Investigators, the IRBs and Regulatory Authorities

The sponsor should report any suspected unexpected serious adverse reactions (SUSARs) and other SAEs subjected to the expedited report to regulatory authorities, investigators and the heads of the study sites in accordance with the laws/regulations in the countries where the study is conducted. Relative to the first awareness of the event by/or further provision to the sponsor or its designee, SUSARs will be submitted to regulatory authorities within 7 days for fatal and life-threatening events and 15 days for other serious events. Similarly, the sponsor will submit expedited reports for other significant safety information considered to substantially affect benefit/risk of the study drug, or continuation of treatment or the study itself. The copies of these expedited report-related documents will be submitted to the IRBs in the study sites.

#### 11.0 STUDY-SPECIFIC COMMITTEES

## 11.1 Independent Adjudication Committee for PML

In the study, the Independent Adjudication Committee for PML established to evaluate the PML risk will be utilized. When any PML risk, which may not be ruled out in a neurologist's examination in accordance with the PML checklists in the Appendix D, will be adjudicated in the Independent Adjudication Committee for PML based on the subject data provided. Detailed procedures should be in accordance with the separately specified written procedure.
#### 12.0 DATA HANDLING AND RECORDKEEPING

The full details of procedures for data handling will be documented in the Data Management Plan. AEs, PTEs, medical history, and concurrent conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Drugs will be coded using the World Health Organization (WHO) Drug Dictionary and Japanese Drug Dictionary.

#### 12.1 CRFs (Electronic and Paper)

Completed (e)CRFs are required for each subject signed the informed consent.

The sponsor or the its designee will provide the study sites with access authority to the eCRF. The sponsor will make arrangements to train appropriate site staff in the use of the eCRF. These forms are used to transmit the information collected in the performance of this study to the sponsor and regulatory authorities. Data will be entered directly to the (e)CRF in Japanese.

Reasons for significant corrections should additionally be included. All new additions are to be made with the date and signature or seal affixed.

The principal investigator will verify accuracy and completeness of the records in the (e)CRF and electrically sign on the applicable pages. Furthermore, the investigator must retain full responsibility for the accuracy and authenticity of all data entered on the (e)CRFs.

The following data will not be recorded directly into the (e)CRFs;

- 1) Laboratory test values (except urine pregnancy test)
- 2) Serum concentrations of MLN0002
- 3) HAHA assessment
- 4) Neutralizing antibody assessment
- 5) CDAI score (including each subscore)
- 6) Adjudication of clinical response/no-response at Week 10 (Visit 5)
- 7) Items of follow-up survey

After the database lock of clinical study database, any change of, modification of or addition to the data on the (e)CRFs should be made by the investigator with use of change and modification records of (e)CRFs (Data Clarification Form) provided by the sponsor. The principal investigator must review the Data Clarification Form for completeness and accuracy, and must sign, or sign and seal, and date the form.

The (e)CRFs will be reviewed for completeness and acceptability at the study site during periodic visits by study monitors. The sponsor or its designee will be permitted to review the subject's medical and hospital records pertinent to the study to ensure accuracy of the (e)CRFs. The completed (e)CRFs are the sole property of the sponsor and should not be made available in any form to third parties, except for authorized representatives of appropriate governmental health or regulatory authorities, without written permission of the sponsor.

#### 12.2 Record Retention

Investigators or the heads of the study sites should retain the following documents in addition to records clearly specified in Section 12.1 and the study-specific documents for inspections or audits by regulatory authorities and the sponsor or its designee. These documents include the subject list for screening, medical records, worksheets for the study, the original informed consents with the signatures/dates, electronic copies of the (e)CRFs including tracking of audit certifications, and the drug control records. In addition, investigators and the heads of the study site should retain the retentive essential documents until the following 1) or 2), whichever comes later. However, when the sponsor requires a longer retention period than the above, the retention period and manner will be discussed among the sponsor and the heads of the study sites.

- 1) The marketing approval day for the drug (when the study was terminated, for 3 years since receipt of the termination notice)
- 2) The same day after 3 years as the study termination or completion day

Furthermore, investigators and the heads of the study sites should retain the retentive essential documents until receipt of the notice stating that these documents should not be retained any more from the sponsor.

#### 13.0 STATISTICAL METHODS

## 13.1 Statistical and Analytical Plans

Since the study has different objectives in the induction phase and maintenance phases/open-label cohort, analyses will be conducted separately among these.

The Statistician in the study will prepare and finalize the Statistical Analysis Plan prior to blind-breaking. The document will provide further details regarding the definition of analysis variables and analysis methodology to address all study objectives.

The double-blinded review should be conducted prior to blind-breaking. In the double-blinded review, accuracy and completeness of the study data, feasibility of subject evaluation, and acceptability of the planned analysis methodology will be evaluated.

The data for marketing application will be analyzed, which includes data of all subjects as fixed on the cut-off date for marketing application. Additionally, the open-label cohort will be analyzed separately at the time when the last subject completed the study.

#### 13.1.1 Analysis Sets

In the study, 3 types of analysis sets will be used in the induction phase, i.e., the "Full Analysis Set of the induction phase," "Per Protocol Set of the induction phase" and "Safety Analysis Set of the induction phase."

The "Full Analysis Set of the induction phase," a primary population for the efficacy analysis in the induction phase, is defined as "subjects who were randomized and received at least one dose of the study drug in the induction phase."

Three types of analysis sets will be used in the maintenance phase, i.e., the "Full Analysis Set of the maintenance phase," "Per Protocol Set of the maintenance phase" and "Safety Analysis Set of the maintenance phase."

The "Full Analysis Set of the maintenance phase," a primary population for the efficacy analysis in the maintenance phase, is defined as "subjects who were randomized and received at least one dose of the study drug in the maintenance phase."

Two types of analysis sets will be used in the open-label cohort, i.e., the "Full Analysis Set in the open-label cohort" and "Safety Analysis Set in the open-label cohort."

The "Safety Analysis Set in the open-label cohort" in the open-label cohort, a population for the safety analysis, is defined as "subjects who received at least one dose of the study drug in the open-label cohort."

The detailed definitions of analysis sets are specified separately in the "Data-Handling Rules for Analyses."

The sponsor will verify acceptability of definition of the analysis sets and the data-handling rules for analyses in consultation with medical specialists before database lock, if needed, and add matters not addressed in the plan for finalization as the "Data-Handling Rules for Analyses."

## 13.1.2 Analysis of Demographics and Other Baseline Characteristics

The major subject backgrounds will be calculated by each "treatment group in the induction phase" and in the consolidated "treatment groups in the induction phase" in the "all subjects randomized in the induction phase."

The major subject backgrounds will be calculated by each "treatment group in the maintenance phase" and in the consolidated "treatment groups in the maintenance phase" in the "all subjects randomized in the maintenance phase."

The major subject backgrounds will be calculated in the "all subjects enrolled into the open-label cohort."

The major subject backgrounds will be calculated in "all subjects who received the placebo in the induction phase and enrolled into the maintenance phase."

#### 13.1.3 Efficacy Analysis

## (1) Primary Endpoint and Analysis Methodology in the Induction Phase

[Primary endpoint]

CDAI-100 response at Week 10

[Primary analysis]

The following descriptive calculations will be performed in the "Full Analysis Set in the induction phase."

"CDAI-100 response at Week 10" (primary endpoint of the induction phase) will be calculated by treatment group of the induction phase. Also clinical response at Week 10 will be calculated with stratification according to a history of anti-TNF $\alpha$  antibody therapy and the comparison will be made with the Cochran-Mantel-Haenszel (CMH) test with 2-sided significance level of 10% by using a history of anti-TNF $\alpha$  antibody therapy as a stratification factor.

The results of the primary analysis of the induction phase will be interpreted as below to determine the efficacy of MLN0002 induction therapy.

• The superiority of MLN0002 over the placebo on CDAI-100 response at Week 10 in the primary analysis of the induction phase is demonstrated when a statistically significant difference is observed in the CDAI-100 response at Week 10.

[Secondary analysis]

For sensitivity point of view, robustness of the results will be confirmed in the same manner as those in the primary analysis described in Section 13.1.3 (1) in the "Per Protocol Set of the induction phase."

## (2) Secondary Endpoints and Analysis methodologies in the Induction Phase

[Secondary endpoints]

Clinical remission at Week 10

Change in CRP level over time in the subpopulation of subjects with the baseline CRP level of >0.30 mg/dL

[Secondary analysis]

Clinical remission at Week 10 will be calculated in the same manner as those in the primary analysis described in Section 13.1.3 (1) in the "Full Analysis Set in the induction phase."

The results of the secondary analysis will be interpreted as below to determine the efficacy of MLN0002 induction therapy.

• The superiority of MLN0002 over the placebo on clinical remission at Week 10 in the primary analysis of the induction phase is demonstrated when a statistically significant difference is observed in both the CDAI-100 response at Week 10 and clinical remission at Week 10.

[Other analyses]

The following analysis will be conducted in subjects with the baseline CRP level of >0.30 mg/dL in the "Full Analysis Set in the induction phase".

Summary statistics of CRP levels measured at each evaluation in the induction phase will be calculated by each treatment group.

Summary statistics of change of CRP level at each evaluation in the induction phase from that at baseline will be calculated by each treatment group.

## (3) Exploratory Endpoints in Induction Phase

See Section 5.2.1.3.

## (4) Primary Endpoint and Analysis Methodology in the Maintenance Phase

[Primary endpoint]

Clinical remission at Week 60

[Primary analysis]

The following descriptive calculations will be performed in the "Full Analysis Set in the maintenance phase."

The "clinical remission at Week 60" (primary endpoint of the maintenance phase) will be calculated by treatment group in the maintenance phase.

[Secondary analysis]

For sensitivity point of view, robustness of the results will be confirmed in the same manner as those in the primary analysis described in Section 13.1.3 (4) in the "Per Protocol Set of the maintenance phase."

#### (5) Secondary Endpoints and Analysis Methodology in the Maintenance Phase

[Secondary endpoints]

CDAI-100 response at Week 60

Durable remission in the maintenance phase

Corticosteroid-free remission at Week 60

[Analysis methodology]

CDAI-100 response at week 60, durable response in the maintenance phase and corticosteroid-free remission at Week 60 will be analyzed in the same manner as those in the primary analysis described in the Section 13.1.3 (4) in the "Full Analysis Set in the maintenance phase".

## (6) Exploratory Endpoints in Maintenance Phase

See Section 5.2.2.3.

#### (7) Data Transformation and Missing Data

Details are specified in the "Data-Handling Rules for Analyses" and the "Statistical Analysis Plan."

In the analysis of the efficacy endpoints of clinical response and clinical remission, when adjudications for these endpoints were missing at the time of evaluation, non-responder and non-remitter will be imputed.

## (8) Significance Level and Confidence Coefficient

• Significance level: 10% (2-sided test)

• Confidence coefficient: 95% (2-sided estimate)

#### 13.1.4 Pharmacokinetic Analysis

[Endpoints]

Serum concentrations of MLN0002

[Analysis methodology]

Summary statistics for serum MLN0002 concentrations at each evaluation in the induction phase will be calculated in the subjects who underwent proper determination of serum MLN0002

concentrations out of the "Full Analysis Set of the induction phase," and subsequently figures showing transition of means/standard deviations will be plotted.

Summary statistics for serum MLN0002 concentrations at each evaluation in the maintenance phase will be calculated in the subjects who underwent proper determination of serum MLN0002 concentrations out of the "Full Analysis Set of the maintenance phase" by each treatment group in the maintenance phase, and subsequently figures showing transition of means/standard deviations will be plotted.

#### 13.1.5 Safety Analysis

## (1) AEs in the induction phase

AEs will be summarized in the "Safety Analysis Set in the induction phase."

Treatment-emergent AEs (TEAEs) in the induction phase are defined as AEs that emerged during the period from the first dose of the study drug in the induction phase through the first dose of the study drug in the maintenance phase or open-label cohort in the subjects enrolled into the maintenance phase or the open-label cohort, or defined as AEs that emerged since the first dose of the study drug in the induction phase in the subjects not enrolled into the maintenance phase or open-label cohort.

The following analyses will be conducted for TEAEs in the induction phase by treatment group in the induction phase. All TEAEs will be coded by use of MedDRA, and summarized based on the System Organ Class and Preferred Term.

- Calculation of overall TEAEs
- Calculation of "study drug-related" TEAEs
- Calculation of overall TEAEs by severity
- Calculation of "study drug-related" TEAEs by severity
- Calculation of TEAEs leading to "dose discontinuation" in disposition.
- Calculation of serious TEAEs
- Calculation of overall TEAEs by start period

#### (2) AEs in the maintenance phase

TEAEs in the maintenance phase are defined as AEs that emerged during the period from the first dose of the study drug in the maintenance phase through the first dose of the study drug in the open-label cohort in the subjects who enrolled into the open-label cohort, or defined as AEs emerged since the first dose of the study drug in the maintenance phase in the subjects not enrolled into the open-label cohort.

TEAEs in the maintenance phase will be analyzed in the same manner as those described in Section 13.1.5 (1) by each treatment group in the maintenance phase in the "Safety Analysis Set of the maintenance phase."

TEAEs in the maintenance phase will be analyzed in the same manner as those described in Section 13.1.5 (1) in "subject allocated to the placebo group in the induction phase and who received the placebo in the maintenance phase."

## (3) AEs in the Open-label Cohort

TEAEs in the open-label cohort are defined as AEs emerged after the first dose of the study drug in the open-label cohort.

TEAEs in the open-label cohort will be analyzed in the same manner as those described in the Section 13.1.5 (1) in the "Safety Analysis Set of the open-label cohort."

## (4) AEs Emerged after Treatment of MLN0002

TEAEs emerged after treatment of MLN0002 are defined as AEs emerged after the first dose of MLN0002.

TEAEs emerged after treatment of MLN0002 will be analyzed in the same manner as those described in Section 13.1.5 (1) in "subjects who received at least one dose of MLN0002."

#### (5) Laboratory tests, 12-Lead ECG, Vital Signs and Body Weights

The analysis sets and groups to be analyzed are the same as those described in (1), (2) and (3) in Section 13.1.5 in principle.

Summary statistics of measured values and difference between pre-/post-treatments will be calculated by each evaluation timing. Figures showing transition of each test value will be plotted.

Shift tables showing difference between pre-/post-treatments will be created.

#### 13.1.6 Analysis of Immunogenicity Endpoints

[Endpoints]

HAHA, neutralizing antibody

[Analysis methodology]

HAHA /neutralizing antibody test results will be calculated in the subjects who underwent proper HAHA /neutralizing antibody test out of the "Full Analysis Set of the induction phase."

HAHA /neutralizing antibody test results will be calculated by each treatment group in the maintenance phase in the subjects who underwent a HAHA /neutralizing antibody test out of the "Full Analysis Set of the maintenance phase."

HAHA /neutralizing antibody test results will be calculated in the subjects who underwent a HAHA /neutralizing antibody test out of the "Full Analysis Set of the open-label cohort."

## 13.2 Interim Analysis and Criteria for Early Termination

The data for marketing application will be analyzed, which includes data of all subjects as fixed on the cut-off date for marketing application. Continuation/termination of the study will not be judged based on the analysis.

#### 13.3 Determination of Sample Size

Subjects to be randomized in the induction phase: 110 to 152 subjects

Number of subjects to be evaluated in the induction phase (number of "subjects randomized and who received at least one dose of the study drug in the induction phase")

MLN0002 group in the induction phase: 55 to 76 subjects

Placebo group in the induction phase: 55 to 76 subjects

Total: 110 to 152 subjects

Subjects to be enrolled into the maintenance phase: approximately 53 to 73 subjects

Number of subjects to be evaluated in the maintenance phase (number of "subjects randomized and who received at least one dose of the study drug in the maintenance phase")

MLN0002 group in the maintenance phase: approximately 16 to 22 subjects

Placebo group in the maintenance phase: approximately 16 to 22 subjects

Total: approximately 32 to 44 subjects

[Justification of the sample size]

On the basis of the findings from the phase 3 double-blinded, placebo-controlled study of MLN0002 in non-Japanese moderate to severe CD subjects who had failed with an anti-TNF $\alpha$  antibody (C13011), the CDAI-100 response at Week 10 in MLN0002 and the placebo was estimated as 47.2% and 24.6%, respectively, clinical remission at Week 10 in MLN0002 and the placebo was estimated as 28.7% and 13.0%, respectively, and the CDAI-70 response at Week 10 in MLN0002 and the placebo was estimated as 56.9 % and 38.7%, respectively, in the study.

When the CDAI-100 response at Week 10 in the induction phase is analyzed using Pearson's chi-square test with 2-sided significance level of 10%, 55 subjects each (at a ratio of 1:1, total 110 subjects) will be required for the MLN0002 and placebo group to detect significance with a power of at least 80%. These numbers were therefore selected as numbers of evaluable subjects of the primary endpoint of the induction phase. When the clinical remission at Week 10 is analyzed in the same manner on the accumulated 55 to 76 subjects to be evaluated for the primary endpoint in the induction phase, statistical significances in both the CDAI-100 response at Week 10 and clinical remission at Week 10 are detected with a power of 61% to 76%...

Number of subjects to be evaluated for the primary endpoint in the maintenance phase will be 16 to 22 subjects in each group and 32 to 44 subjects in total, when such results are obtained as estimated in the above.

## 14.0 QUALITY CONTROL AND QUALITY ASSURANCE

## 14.1 Study-Site Monitoring Visits

Monitoring visits to the study site will be made periodically during the study to ensure that all aspects of the protocol are followed. Source documents will be reviewed for verification of data recorded on the (e)CRFs. Source documents are defined as original documents, data, and records. The investigator and head of the study site should assure the sponsor (or its designee) or the IRB to review source documents.

The sponsor or its designee will review records including Investigator's files, drugs, subjects' medical records and informed consents to verify that the study is being conducted properly in compliance with the protocol. In addition, consistency will be verified between raw data and the (e)CRF. It is important that the investigator and other study personnel are available during the monitoring visits and that sufficient time is devoted to the process.

#### 14.2 Protocol Deviations

Investigators may deviate from or modify the protocol without prior written agreement with the sponsor and prior approval from the IRB in medically inevitable occasions including any danger in subjects to be avoided urgently. After that, the investigator will give notice about details and reasons of the deviation or modification to the sponsor and the head of the study site in writing, retaining a copy, and discuss revisions of the protocol with the sponsor for agreement, if needed. If revision is needed, a draft of the revision will be submitted to the head of the study site at the earliest possible time to be approved by the IRB.

Investigators will record all deviations from the protocol.

#### 14.3 Quality Assurance Audits and Regulatory Agency Inspections

The study site also may be subject to quality assurance audits by the sponsor or designees. In this circumstance, the sponsor-designated auditor will contact the site in advance to arrange an auditing visit. The auditor may ask to visit the facilities where laboratory samples are collected, where the drug is stored and prepared, and any other facility used during the study. In addition, there is the possibility that this study may be inspected by regulatory agencies, including those of foreign governments (e.g., the FDA, the United Kingdom Medicines and Healthcare products Regulatory Agency). If the study site is contacted for an inspection by a regulatory body, the sponsor should be notified immediately. The Investigator and the head of institution guarantee access for quality assurance auditors to all study documents as described in Section 14.1.

#### 15.0 ETHICAL ASPECTS OF THE STUDY

This study will be conducted with the highest respect for the individual participants (i.e., subjects) according to the protocol, the ethical principles that have their origin in the Declaration of Helsinki, and the ICH Harmonised Tripartite Guideline for GCP. Each Investigator will conduct the study according to applicable local or regional regulatory requirements and align his or her conduct in accordance with the "Responsibilities of the Investigator" that are listed in Appendix B.

## 15.1 IRB Approval

IRBs will be established in accordance with local laws/regulations in the area where the study will be conducted. The sponsor or its designee will obtain a document describing names and titles of members of the IRB If any member of the IRB directly participates in this study, written notification regarding his or her abstinence from voting must also be obtained.

The sponsor or designee will supply relevant documents for submission to the respective IRB for the protocol's review and approval. This protocol, Investigator's Brochure, a copy of the informed consent form, and, if applicable, subject recruitment materials and/or advertisements and other documents required by all applicable laws and regulations, must be submitted to a central or local IRB for approval. The sponsor or its designee will obtain an approval document for the protocol and the informed consent form the IRB prior to the first dose of the study (i.e., before delivery of sponsor-supplied drugs). The IRB approval must refer to the study by exact protocol title, number, and version date; identify versions of other documents (e.g., informed consent form) reviewed; and state the approval date. The drugs will be dispatched after sponsor's validation of regulatory documents in the study site. Any procedures in the screening phase described in the protocol should not be started until the study site receives the drugs.

The study site should comply with all requirements specified by the IRB. This may include notification to the IRB regarding protocol amendments, updates to the informed consent form, recruitment materials intended for viewing by subjects, local safety reporting requirements, reports and updates regarding the ongoing review of the study at intervals specified by the respective IRB, and submission of the Investigator's final status report to the IRB. All IRB approvals and relevant documentation for these items must be provided to the sponsor or its designee.

Subject incentives should not exert undue influence for participation. Subject incentives should be approved by the IRB and the sponsor.

Regarding pharmacogenomic investigation using collected and stored specimens, analysis will be carried out at the time when detail is determined. The sponsor will create a research protocol for pharmacogenomics investigations and a research protocol will require prior approval of the company IRB in Japan.

#### 15.2 Subject Information, Informed Consent, and Subject Authorization

Written consent documents will embody the elements of informed consent as described in the Declaration of Helsinki and the ICH Guidelines for GCP and will be in accordance with all **CONFIDENTIAL** 

applicable laws and regulations. Written consent documents describe availability and disclosure (to any third-parties inside/outside Japan) of subjects' personal information and personal medical information in the study. The informed consent includes detailed explanation pertaining to primary intention, purpose, and possible risks/benefits. The informed consent form will detail the requirements of the participant and the fact that he or she is free to withdraw at any time without giving a reason and without prejudice to his or her further medical care.

Investigators have responsibility for preparation, contents and approval to be obtained from the IRB for the informed consent. The informed consent should be approved by the IRB prior to being effective.

The informed consent should be described in understandable wording for subjects. Investigators must explain the contents of the informed consent thoroughly to the subjects. Information should be provided in a proper manner as approved by the IRB both orally or in writing, where possible. In the event the subject is not capable of rendering adequate written informed consent, then the subject's legally acceptable representative may provide such consent for the subject in accordance with applicable laws and regulations.

The subject, or the subject's legally acceptable representative, must be given ample opportunity to: (1) inquire about details of the study and (2) decide whether or not to participate in the study. The subject or the subject's legally acceptable representative, when he/she has decided to participate in the study, should enter the signature (or name/seal) and date on the informed consent prior to participation. Investigators should request the subject or the subject's legally acceptable representative to enter his/her formal (not nicknames, etc.) signature or name/seal by use of a black or blue ballpoint pen. Investigators should enter the signature (or name/seal) and date on the informed consent prior to the subject's participation in the study, as well.

Investigators should retain originals of the informed consent with signatures or names/seals. Investigators should record the date of acquisition of the subject's signature or name/seal on the informed consent in the subject's medical record. Additionally, a copy of the informed consent with the signatures or names/seals will be provided to the subject.

All revised informed consent forms must be reviewed and signed by relevant subjects or the relevant subject's legally acceptable representative in the same manner as the original informed consent. The date the revised consent was obtained should be recorded in the subject's medical record, and the subject should receive a copy of the revised informed consent form.

The Pharmacogenomic Research will be explained based on "the informed consent for the Pharmacogenomic Research in the study for MLN0002" to the subjects who were given an explanation by use of the informed consent of the study. Sampling for Pharmacogenomic Research will be performed in the subjects who gave both informed consents for the study and the pharmacogenomic investigation.

When a subject requests disposal of his/her retained samples, it will be implemented according to Section 9.4.

## 15.3 Subject Confidentiality

The sponsor and designees affirm and uphold the principle of the subject's right to protection against invasion of privacy. Throughout this study, a subject's source data will only be linked to the sponsor's clinical study database or documentation via a unique identification number. As permitted by all applicable laws and regulations, limited subject attributes, such as sex, age, or date of birth may be used to verify the subject and accuracy of the subject's unique identification number.

To comply with ICH Guidelines for GCP and to verify compliance with this protocol, the sponsor requires the investigator to permit its monitor or designee's monitor, representatives from any regulatory authority (e.g., FDA, Medicines and Healthcare products Regulatory Agency, Pharmaceuticals and Medical Devices Agency), the sponsor's designated auditors, and the appropriate IRBs to review the subject's original medical records (source data or documents), including, but not limited to, laboratory test result reports, ECG reports, admission and discharge summaries for hospital admissions occurring during a subject's study participation, and autopsy reports. Access to a subject's original medical records requires the specific authorization of the subject as part of the informed consent process (see Section 15.2).

Copies of any subject source documents that are provided to the sponsor must have certain personally identifiable information removed (i.e., subject name, address, and other identifier fields not collected on the subject's [e]CRF).

## 15.4 Publication, Disclosure, and Clinical Trial Registration Policy

#### 15.4.1 Publication and Disclosure

The investigator is obliged to provide the sponsor with complete test results and all data derived by the investigator from the study. During the study, only the sponsor may make study information available to other study investigators or to regulatory agencies, except as required by law or regulation. Except as otherwise allowable in the clinical study site agreement, any public disclosure (including publicly accessible websites) related to the protocol or study results is the sole responsibility of the sponsor.

The sponsor may publish any data and information from the study (including data and information generated by Investigators) without the consent of investigators.

The investigator, when intends to publicly present information acquired in the course of the study at a specialized academic society, etc., should obtain prior written approval from the sponsor.

#### 15.4.2 Clinical Trial Registration

In order to ensure that information on clinical trials reach the public in a timely manner and to comply with applicable law, regulation and guidance, Takeda will, at a minimum, register all clinical trials conducted in subjects that it sponsors anywhere in the world on ClinicalTrials.gov or other publicly accessible websites (including JAPIC-CTI) before trial initiation. Takeda contact

information, along with Investigator's city, state (for US investigators), country, and recruiting status will be registered and available for public viewing.

#### 15.4.3 Clinical Trial Results Disclosure

Takeda will post the results of this clinical trial, regardless of outcome, on ClinicalTrials.gov or other publicly accessible websites (including JAPIC-CTI), as required by applicable laws and/or regulations.

#### 15.5 Insurance and Compensation for Injury

Any health damage occurred in subjects participating in the study will be compensated according to the local regulation applied to the study site. The sponsor or its designee will insure subjects be compensated for health damage, when required in the area where the study is conducted.

Subjects suffering/suffered health damage will be compensated in accordance with the study contract. Investigators will contact the sponsor or its designee for any questions pertaining to compensation.

#### 16.0 REFERENCES

- [1] Diagnostic Criteria and Treatment Guideline for Ulcerative Colitis and Crohn's Disease. "Research Group for Intractable Inflammatory Bowel Disease" Designated as Specified Disease by the MHLW of Japan (the Group of Dr. Watanabe), the additional volume of Assigned Study Report in 2012.
- [2] Soler D, Chapman T, Yang LL, Wyant T, Egan R, Fedyk ER. The binding specificity and selective antagonism of vedolizumab, an anti-alpha4beta7 integrin therapeutic antibody in development for inflammatory bowel diseases. J Pharmacol Exp Ther. 2009;330:864-75.
- [3] Edula RG, Picco MF. An evidence-based review of natalizumab therapy in the management of Crohn's disease. Ther Clin Risk Manag. 2009;5:935-42.
- [4] Tilg H, Kaser A. Vedolizumab, a humanized mAb against the α4β7 integrin for the potential treatment of ulcerative colitis and Crohn's disease. Curr Opin Investig Drugs. 2010;11:1295-304.
- [5] Parikh A, Leach T, Wyant T, Scholz C, Sankoh S, Mould DR, et al. Vedolizumab for the treatment of active ulcerative colitis: A randomized controlled phase 2 dose-ranging study. Inflamm Bowel Dis. 2012;18:1470-9.
- [6] Feagan BG, Greenberg GR, Wild G, Fedorak RN, Paré P, McDonald JW, et al. Treatment of ulcerative colitis with a humanized antibody to the alpha4beta7 integrin. N Engl J Med. 2005;352:2499-507.
- [7] Feagan BG, Greenberg GR, Wild G, Fedorak RN, Paré P, McDonald JW, et al. Treatment of active Crohn's disease with MLN0002, a humanized antibody to the alpha4beta7 integrin. Clin Gastroenterol Hepatol. 2008;6:1370-7.
- [8] Feagan BG, Rutgeerts P, Sands BE, Hanauer S, Colombel JF, Sandborn WJ, et al. Vedolizumab as induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2013;369(8):699-710.
- [9] Sandborn WJ, Feagan BG, Rutgeerts P, Hanauer S, Colombel JF, Sands BE, et al. Vedolizumab as induction and maintenance therapy for Crohn's disease. N Engl J Med. 2013; 369(8):711-21.
- [10] Sands B; Feagan B, Rutgeerts P, Colombel J; Sandborn W; Sy R, et al. Vedolizumab induction therapy for patients with Crohn's disease and prior anti-TNF failure: a randomized, placebo-controlled, double-blind, multicenter trial. Presented at: Crohn's & Colitis Foundation of America Advances in Inflammatory Bowel Diseases Clinical and Research Conference. December 13-15, 2012. Hollywood, FL.
- [11] Kobayashi K, Suzuki Y, Watanabe K, Mukae M, Yamada T, Yamagami H. The phase I, multicenter, open-label, dose-escalation, repeated-dose study for VDZ in Japanese CD patients. The 21st Japan Digestive Disease Week, Tokyo, 2013.

- [12] Kappos L, Bates D, Edan G, Eraksoy M, Garcia-Merino A, Grigoriadis N, et al. Natalizumab treatment for multiple sclerosis: updated recommendations for patient selection and monitoring. Lancet Neurol. 2011;10:745-58.
- [13] Best W.R., Backtel J.M., Singleton J.W., et al.: Development of Crohn's disease activity index. Gastroenterology 1976;70:439-444.

# Appendix A Schedule of Study Procedures

## Screening, Induction Phase, Maintenance Phase

| | | Screening | | Indu | ction F | Phase | | | | | | Ma | intena | nce Ph | ase | | | | | 16 weeks | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Week <sup>a</sup> | | 0 | 2 | 6 | 10/ET <sup>j</sup> | 14 | 18 | 22 | 26 | 30 | 34 | 38 | 42 | 46 | 50 | 54 | 58 | 60/ETk | after the | led |
| Study | Day <sup>a</sup> | -21 to -7i | 1 | 15 | 43 | 71/ET <sup>j</sup> | 99 | 127 | 155 | 183 | 211 | 239 | 267 | 295 | 323 | 351 | 379 | 407 | 421/ETk | last dose | g <u>.</u> |
| Procedures | Visit Windows (Days) a | _ | _ | ±3 | ±3 | ±3/ET <sup>j</sup> | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | -7 - +6 | ±7/ET <sup>k</sup> | ±14 | Unscheduled<br>visits <sup>1</sup> |
| | Visit | 1 | 2 | 3 | 4 | 5/ET <sup>j</sup> | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18/ET <sup>k</sup> | - | |
| Informed cons | sent | X | | | | | | | | | | | | | | | | | | | |
| Inclusion/excl | usion criteria | X <sup>m</sup> | X | | | | | | | | | | | | | | | | | | |
| Demographics<br>medical histor<br>complications | y, prior therapies, | X <sup>m</sup> | | | | | | | | | | | | | | | | | | | |
| Randomizatio | n | | X | | | | X | | | | | | | | | | | | | | |
| Issuance of stu<br>numbers/admi | | | X | X | X | | X | | X | | X | | X | | X | | X | | | | |
| Physical exam | ination, vital signs <sup>b</sup> | Xm | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Body weight <sup>b</sup> | | Xm | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ECG <sup>b</sup> | | Xm | X | | | X | | | | | | | | | | | | | X | X | |
| Chest Imaging | g Procedure <sup>c</sup> | X <sup>m</sup> | | | | | | | | | | | | | | | | | | X | |
| Tuberculosis 7 | Γest | Xn | | | | | | | | | | | | | | | | | | | |
| PML checklist | ts <sup>b</sup> | Xm | X | X | X | | X | | X | | X | | X | | X | | X | | | X | |
| ے Blood b | iochemistry | Xn | X | X | X | X | X | | X | | X | | X | | X | | X | | X | X | |
| Hemato | | Xn | X | X | X | X | X | | X | | X | | X | | X | | X | | X | X | |
| Urinaly | | X <sup>n</sup> | X | | | X | X | | | | | | | | | | | | X | X | |
| 턴 Urine p | regnancy test <sup>d</sup> | Xm | X | X | X | X | X | | X | | X | | X | | X | | X | | X | X | |
| | tigen, HCV antibody,<br>tigen/antibody | X <sup>n</sup> | | | | | | | | | | | | | | | | | | | |
| inflamn | natory markers | Xn | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | |
| CDAI score | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Blood samplin | ng for hematocrit teste | | X | (X) | (X) | X | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | | (X) |
| Check of the p | atient diary | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| IBDQ <sup>b</sup> | | | X | | | X | X | | | | | | X | | | | | | X | | |
| Blood samplin<br>HAHA/neutra | ng for<br>lizing antibody test <sup>f</sup> | | X | | | X | | | | | X | | | | | | | | X | X | |
| Blood samplin | ng for PK <sup>f</sup> | | | X | X | X | X | | X | | X | | | | | | | | X | | |
| Blood samplin | | | X | | | | | | | | | | | | | | | | | | |
| Concomitant of | lrug/therapy | X <sup>m</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PTEs/AEsh | | X <sup>m</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

Footnotes are on last table page.

# Appendix A Schedule of Study Procedures (continued)

## **Open-label Cohort**

| | | | | | | | | Open-lab | el Cohort | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Week <sup>a</sup> | 0x | 2x | 6x | 10x | 14x | 18x | 22x | 26x | 30x | 34x | 38x | 42x | 46x | 50x |
| Study | Day <sup>a</sup> | 1x | 15x | 43x | 71x | 99x | 127x | 155x | 183x | 211x | 239x | 267x | 295x | 323x | 351x |
| Procedures | Visit Windows<br>(Days) <sup>a</sup> | _ | ±3 | ±3 | ±3 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 |
| | Visit | 1x | 2x | 3x | 4x | 5x | 6x | 7x | 8x | 9x | 10x | 11x | 12x | 13x | 14x |
| Informed conse | ent | | | | | | | | | | | | | | |
| Inclusion/exclu | | | | | | | | | | | | | | | |
| Demographics,<br>medical history<br>complications | body height,<br>, prior therapies, | | | | | | | | | | | | | | |
| Randomization | | | | | | | | | | | | | | | |
| Issuance of stu-<br>numbers/admin | | $X^q$ | X | X | | X | | X | | X | | X | | X | |
| Physical exami | nation, vital signs <sup>b</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Body weight <sup>b</sup> | | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ECG <sup>b</sup> | | | | | | | | | | | | | | | |
| Chest Imaging | Procedure <sup>c</sup> | | | | | | | | | | | | | | |
| Tuberculosis T | est | | | | | | | | | | | | | | |
| PML checklists | sb | $X^q$ | X | X | | X | | X | | X | | X | | X | |
| | iochemistry | | X | X | | X | | X | | X | | X | | X | |
| Hemato | logy | | X | X | | X | | X | | X | | X | | X | |
| Urinaly: | | | | | | | | | | | | | | | |
| Urine p | regnancy test <sup>d</sup> | | X | X | | X | | X | | X | | X | | X | |
| HBs ant | rigen, HCV antibody,<br>rigen/antibody | | | | | | | | | | | | | | |
| Inflamn | natory markers | | X | X | | X | | X | | X | | X | | X | |
| CDAI score | | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Blood sampling | g for hematocrit teste | | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) |
| Check of the pa | ntient diary | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| IBDQ <sup>b</sup> | | | | | | | | | | | | | | | |
| | izing antibody testf | | | | X | | | | | X | | | | | |
| Blood sampling | | | | | | | | | | | | | | | |
| Blood sampling | | | | | | | | | | | | | | | |
| Concomitant di | rug/therapy | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PTEs/AEsh | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

Footnotes are on last table page.

## Appendix A Schedule of Study Procedures (continued)

#### **Open-label Cohort (continued)**

| | | _ | | | | | Оро | en-label C | Cohort | | | | | 16 weeks | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| G. | | Week <sup>a</sup> | 54x | 58x | 62x | 66x | 70x | 74x | 78x | 82x | 86x | 90x | 94x/ET <sup>p</sup> | after the last | |
| | udy<br>edures | Day <sup>a</sup> | 379x | 407x | 435x | 463x | 491x | 519x | 547x | 575x | 603x | 631x | 659x/ET <sup>p</sup> | dose | Unscheduled<br>visits <sup>1</sup> |
| rioce | euures | Visit Windows (Days) a | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7/ET <sup>p</sup> | ±14 | VISIUS |
| | | Visit | 15x | 16x | 17x | 18x | 19x | 20x | 21x | 22x | 23x | 24x | 25x/ET <sup>p</sup> | _ | |
| | d consent | | | | | | | | | | | | | | |
| | | on criteria | | | | | | | | | | | | | |
| Demogra | aphics, b | ody height, medical history, | | | | | | | | | | | | | |
| | | omplications | | | | | | | | | | | | | |
| Random | ization | | | | | | | | | | | | | | |
| | | drug numbers/administration | X | | X | | X | | X | | X | | Xr | | |
| Physical | examina | tion, vital signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| Body we | eight <sup>b</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ECG <sup>b</sup> | | | | | | | | | | | | | X | X | |
| Chest In | naging Pr | ocedure <sup>c</sup> | | | | | | | | | | | | X | |
| Tubercu' | losis Tes | t | | | | | | | | | | | | | |
| PML che | ecklists <sup>b</sup> | | X | | X | | X | | X | | X | | X | X | |
| ф | Blood b | oiochemistry | X | | X | | X | | X | | X | | X | X | |
| Laboratory tests <sup>b</sup> | Hemato | logy | X | | X | | X | | X | | X | | X | X | |
| / te | Urinaly | sis | | | | | | | | | | | X | X | |
| ory | Urine p | regnancy test <sup>d</sup> | X | | X | | X | | X | | X | | X | X | |
| orat | | tigen, HCV antibody, | | | | | | | | | | | | | |
| apc | | tigen/antibody tests | | | | | | | | | | | | | |
| Ĺ | Inflamn | natory markers | X | | X | | X | | X | | X | | X | | |
| CDAI sc | core | · | X | X | X | X | X | X | X | X | X | X | X | | X |
| Blood sa | ampling f | or hematocrit teste | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | | (X) |
| | f the pati | | X | X | X | X | X | X | X | X | X | X | X | | X |
| IBDQ <sup>b</sup> | | Ĭ | | | | | | | | | | | | | |
| Blood sa | mpling f | or HAHA/neutralizing | | | 37 | | | | | | | | 37 | 37 | |
| antibody | | Ü | | | X | | | | | | | | X | X | |
| | ampling f | or PK <sup>f</sup> | | | | | | | | | | | | | |
| Blood sa | impling f | for PGx <sup>f</sup> | | | | | | | | | | | | | |
| | | g/therapy | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PTEs/AI | | | X | X | X | X | X | X | X | X | X | X | X | X | X |

ET=early termination, PK=pharmacokinetics, IBDQ=Inflammatory Bowel Disease Questionnaire, HAHA=human anti-human antibody, PTE=pretreatment event


a. The date of the first dose of the study drug in the induction phase is Week 0 (Day 1). The acceptable time windows are given as the number of days away from each scheduled visit.

b. Will be performed before administration of the study drug on the day of study drug administration.

- c. Not required when a chest image performed within 3 months is available (the image taken before the informed consent date is acceptable at screening).
- d. Will be performed only in women of childbearing potential.
- e. It should be performed on VISITs for CDAI score evaluation for calculation of the CDAI score. If the determination result on the evaluation day is impossible to be obtained, instead the blood sampling result within 14 days before evaluation may be used. It should be performed on VISITs for CDAI score evaluation [indicated as (X)] for calculation of the CDAI score, where possible. However, if the determination result on the evaluation day is impossible to be obtained, the blood should not be sampled and the latest determination result may be used for calculation instead.
- f. If the study drug is administrated in the visit, a blood sample should be drawn immediately before study drug administration. If the study drug is not administrated in the visit, a blood sample can be drawn at any time at visits. All blood sampling will be conducted only in study sites with a cooled centrifuge.
- g. Will be collected only in patients who have consented to participate in PGx research once at the earliest possible time between Visit 2 and study completion.
- h. A PTE is an event that occurred before the first dose of the study drug. An AE is an event that occurred after the first dose of the study drug.
- i. If patients with a history of tuberculosis or those with suspicion of it start preventive isoniazid treatment before study enrollment, screening can be conducted between Day -28 and Day-7. Study drug administration must be conducted 21 or more days after isoniazid administration starts.
- j. Patients who will prematurely withdraw from the study in the induction phase after receiving at least one dose should visit the clinical site and have examinations for discontinuation as soon as possible.
- k. Patients who will prematurely withdraw from the study in the maintenance phase should visit the clinical site and have examinations for discontinuation as soon as possible. Eligible patients will be enrolled into open-label cohort 3 to 9 weeks after the last dose of the study drug in the maintenance phase.
- 1. An unscheduled visit will be made due to worsening of CD, etc. Additional tests will be performed as required.
- m. Can be conducted between Day -21 and Day -1. If patients with a history of tuberculosis or those with suspicion of it start preventive isoniazid treatment before study enrollment, screening can be conducted between Day -28 to Day -1. Study drug administration must be conducted 21 or more days after isoniazid administration starts.
- n. The test results should be obtained by Visit 2.
- o. The date of the enrollment into open-label cohort is Week 0x (Day 1x) and the study site visit on Day 1x is Visit 1x. The acceptable time windows are given as the number of days away from each scheduled visit.
- p. Patients who will prematurely withdraw from the study in the open-label cohort should visit the clinical site and have examinations for discontinuation as soon as possible. And the same examination will be conducted in the study termination scheduled 46 weeks after the last subject will be enrolled into open-label cohort.
- q. Will be performed after enrollment into open-label cohort.
- r. Will not be performed in patients who prematurely withdraw from the study.

## Appendix B Responsibilities of the Investigator

- 1. Execute the study properly as complying with the protocol and GCP in consideration of human rights, safety and welfare of subjects.
- 2. In order to assign some important study-related practices to subinvestigators or study collaborators, prepare lists of the assignments and persons in charge to be submitted to the head of the study site and obtain approval.
- 3. Prepare the informed consent form and revise it, when needed.
- 4. Verify the contents in the study contract.
- 5. Provide sufficient information about the protocol, drugs and individual assignments to subinvestigators and study collaborators, instruct and supervise them.
- 6. Select eligible subjects to the protocol, provide explanations to them in writing, and obtain the written informed consents from them.
- 7. Take responsibility for any study-related medical judgment.
- 8. Assure subjects receive sufficient medical care together with the head of the study site for any study-related clinically-relevant AEs throughout the participation and the subsequent period.
- 9. For a subject being treated in other institutions or other departments, provide information in writing of study participation and completion/withdrawal of the subject to the institution or the physician in other department upon subject's approval, which should be documented.
- 10. Report any occasion requiring expedited reports including SAEs to the head of the study site and the sponsor immediately in writing.
- 11. Decide necessity for opening the emergency key of the particular subject in emergency situation.
- 12. Complete the (e)CRFs accurately and completely with the e-signature to be submitted to the sponsor.
- 13. Check, verify and e-sign (e)CRFs entered by subinvestigators or transcribed from raw data by study collaborators to be submitted to the sponsor.
- 14. Be consulted for revision of the protocol or the like, when proposed by the sponsor
- 15. Report study completion to the head of the study site in writing.

## Appendix C Diagnostic Criteria for CD (Revised on January 17, 2013)

#### 1. Overview

Crohn's Disease (CD) is a granulomatous inflammatory disease of unknown etiology but may be contributed by immune disorder, etc. It is most commonly found in young people with edema or ulcers that emerged primarily in the small or large intestine, leading to development of characteristic conditions such as intestinal stenosis or fistula. The original article described that it is an inflammation of the terminal ileum, however, today, the disease is known to occur in any part of the gastrointestinal tract from the mouth through to the anus. As various complications may be induced even outside the gastrointestinal tract, the disease should be treated as a systemic disease. While clinical manifestation may vary depending on affected sites or extent, gastrointestinal condition including diarrhea or abdominal pain, systemic condition including fever, weight loss or malnutrition, and also complication-induced condition including anemia, arthritis, iritis or skin lesions may emerge. Disease condition and lesions may progress with repetition of recurrence and remission, and often become resistant to treatments to deteriorate social activity.

## 2. Major Concepts

- (1) Most Common Onset Ages: from the late 10s to 20s
- (2) Most Common Sites: mostly either of the small or large intestine or both showing lesions including longitudinal ulcers or a cobblestone appearance.
- (3) Clinical Symptoms: abdominal pain, diarrhea, weight loss or fever are commonly observed. The disease may sometimes emerge as intestinal obstruction, intestinal fistula (internal or external fistula), intestinal perforation or major bleeding, or may emerge as anal lesion-induced symptoms, fever of unknown origin, arthritis or the like without abdominal symptoms (or with unidentified complaint in the abdomen in a few cases).
- (4) Clinical Findings
- A. Lesions in the gastrointestinal tract
- [1] The intestine: longitudinal ulcers <Note 1>, cobblestone appearance <Note 2>, discontinuous or skip lesions, irregular-to-round shaped ulcers, or multiple aphtha <Note 3>
- [2] The anus: anal fissure, cavitating ulcers <Note 4>, intractable anal fistula, perianal abscess, edematous skin tag, anal stenosis, etc.
- [3] The stomach and duodenum: multiple aphtha, irregular-shaped ulcers, bamboo-joint-like appearance, notch-like depression, cobblestone appearance, etc.
- [4] Complications: intestinal stenosis, intestinal obstruction, internal fistula (fistula between the intestine intestine, the intestine bladder, the intestine vagina, etc.), external fistula (fistula between the intestine skin), or malignancy (intestinal cancer or anal fistula cancer)

- B. Lesions outside the gastrointestinal tract (including secondary complications)
- [1] The blood: anemia, hypercoagulability, etc.
- [2] The joints: arthritis enteropathic, ankylosing spondylitis, etc.
- [3] The skin: oral aphtha, erythema nodosum, pyoderma gangrenosum, erythema multiforme exudativum, etc.
- [4] The eyes: iritis, uveitis, etc.
- [5] The nutrient metabolism: growth disorder, hypoproteinemia, trace element deficiency, vitamin deficiency, bone disorder, etc.
- [6] Other: primary sclerosing cholangitis, vasculitis, pancreatitis, cholelithiasis, urolithiasis, hepatic disorder, amyloidosis, etc.
- (5) Findings in laparotomies

Induration longitudinally aligned on the mesenteric side, marked creeping fat, circumferential induration on the intestinal wall, shortening of the intestine, intestinal stenosis, fistulation (internal or external fistulas), intestinal massive adhesion, mesenteric lymphadenopathy, etc., may be observed.

- (6) Pathological Findings
- A. Macroscopic findings on resected specimens
- [1] Longitudinal ulcers <Note 1>
- [2] Cobblestone appearance <Note 2>
- [3] Fistula
- [4] Stenosis
- [5] Irregular-to-round shaped ulcers or aphtha <Note 3>
- B. Histological findings on resected specimens
- [1] Noncaseating epithelioid granuloma (may be found in the local lymph nodes as well) <Note 5>
- [2] Full thickness inflammation <Note 6>
- [3] Local or disproportional inflammation
- [4] Fissure
- [5] Ulcers
- C. Histological findings on the biopsy
- [1] Noncaseating epithelioid granuloma <Note 5>
- [2] Disproportional inflammation

- <Note 1> Ulcers of ≥4 to 5 cm in length commonly, aligned longitudinally along the intestine. The finding may be found in intestinal ischemic lesions or infectious enteritis, but these have different development or clinical courses and are rarely associated with inflammatory polyposis or a cobblestone appearance. Also, the finding may be found in UC, but it shows UC-specific findings in the surrounding mucosa.
- <Note 2> Aggregation of different sizes of protrusions on the mucosa between longitudinal ulcers and the surrounding small ulcers The finding may rarely be observed in intestinal ischemic lesions, but these have a shorter protrusion in height with more remarkable redness.
- <Note 3> These may align longitudinally in the disease.
- <Note 4> Deep and wide painful ulcers in the area from the anal canal to the lower rectum.
- <Note 5> It may also be observed in intestinal tuberculosis, etc.
- <Note 6> It is expansion of inflammation into full thickness of the wall of the gastrointestinal tract primarily due to aggregated lymphocytes

## 3. Diagnostic Criteria

- (1) Primary Findings
- A. Longitudinal ulcers <Note 7>
- B. Cobblestone appearance
- C. Noncaseating epithelioid granuloma <Note 8>
- (2) Secondary Findings
- a. Extensive irregular-to-round shaped ulcers or aphtha in the gastrointestinal tract <Note 9>
- b. The characteristic anal lesions <Note 10>
- c. The characteristic gastroduodenal lesions <Note 11>

#### Definitive patients:

- [1] Patients with A or B in the primary findings <Note 12>
- [2] Patients with C in the primary findings and a or b in the secondary findings
- [3] Patients with all of a, b and c in the secondary findings

#### Suspected patients:

[1] Patients with C in the primary findings and c in the secondary findings


- [2] Patients with A or B in the primary findings, however, in whom UC, intestinal Behcet's disease, simple ulcers or intestinal ischemic lesions may not be ruled out
- [3] Patients only with C in the primary findings < Note 13>
- [4] Patients only with any 2 or 1 in the secondary findings
- < Note 7> These, if in the small intestine, commonly emerge in the mesenteric side
- <Note 8> Diagnosis may be improved with the serial section, and preferably should be judged by a skilled pathologist in the gastrointestinal tract
- <Note 9> These may typically align longitudinally but sometimes may not, and should constantly exist for ≥3 month. Additionally, intestinal tuberculosis, intestinal Behcet's disease, simple ulcers, NSAIDs-induced ulcers, infectious enteritis should be ruled out.
- <Note 10> These include anal fissure, cavitating ulcers, anal fistula, perianal abscess or edematous skin tag, and preferably should be diagnosed by a specialist in proctology with knowledge of CD with reference to the Atlas for Macroscopic Findings of Anal Lesions in CD.
- <Note 11> These include a bamboo-joint-like appearance or notch-like depression, and preferably should be diagnosed by a skilled specialist in CD.
- <Note 12> In patients showing only longitudinal ulcers, intestinal ischemic lesions or UC should be ruled out. In patients showing only a cobblestone appearance, intestinal ischemic lesions should be ruled out.
- <Note 13> Granulomatous inflammatory diseases including intestinal tuberculosis should be ruled out.

## 4. Types of the Disease

The disease is classified into the small intestine type, large intestine type or small/large intestine type based on the existing site of longitudinal ulcers, a cobblestone appearance or stenosis. Patients without these findings or patients with these findings only in rare sites will be classified as the atypical type. The atypical type includes the multiple aphtha type, the cecum/appendix-localized type, the rectum type, the gastroduodenal type.

The disease patterns include the inflammation type without complications, the fistula-forming type, and the stenosis type with stenotic lesions.

[Subjoinder] Indeterminate colitis

A patient, who is difficult to be definitively diagnosed as showing clinical and pathological characteristics of both CD and UC, may come to show more specific findings of either disease in the course of follow-up.

# 5. Classification by Severity

Upon treatment, severity should be classified with reference to the following.

| | CDAI# | Concurrent medical conditions | Inflammation<br>(CRP level) | Treatment Response |
|---|---|---|---|---|
| Mild | 150-220 | None | Small elevation | |
| Moderate | 220-450 | No overt complications including intestinal obstruction, etc. | Overt elevation | No response to treatment for mild cases |
| Severe | 450< | Intestinal obstruction, abscess, etc. | Notable elevation | Poor response to the treatment |

<sup>#:</sup> CDAI (Crohn's disease activity index)

## Appendix D PML Checklists

- The PML checklists will be utilized in visits specified in the protocol, or for a subject complaining such symptoms.
- The purpose of the PML checklists is to identify any obvious neurological changes in a subject since the last evaluation.
- When any subjective symptoms were identified, the corresponding tests to see objective findings should be performed. Any symptoms/findings found on the checklists should be recorded as AEs.
- Subjects should be instructed to visit a neurologist, when any obvious neurological changes were observed. Examinations including MRI using a contrast agent should be performed for collection of information supporting the neurological change, if needed.
- Any positive subjective symptoms or positive objective findings should be provided to the sponsor immediately.

## **Algorithm for Subject Evaluation**



**CONFIDENTIAL** 

# Subjective PML checklist

| Date: | month/ | date/ | year |
|---------|------------|---------|------|
| Subject | Identifica | tion Co | de: |

| Symptoms | Have you had<br>significantly to<br>experience fo<br>following? | unusual | If "yes," describe symptoms specifically | Objective test to be applied: results should be recorded in the Objective PML checklist |
|---|---|---|---|---|
| | Yes | No | | |
| 1. Have you experienced continuous loss of vision, multiple vision or reading disorder, recently? | | | | Visual field and eye movement should be tested. |
| 2. Have you felt any continuous difficulty in talking, or continuous inability of your speech to be understood by others, recently? | | | | Natural observation should<br>be performed for patient's<br>speech for dysarthria or<br>aphasia. The patient should<br>be requested to answer<br>names of some objects and<br>to repeat some phrases<br>with several words. |
| 3. Have you felt any continuous muscle weakness in your arms or legs, recently? | | | | Pronator deflection test (Barré procedure) and/or a test to see ability to keep the arm being rotated Ability to hop on one foot; to tap with the foot and finger. A symmetry test in the muscle. |
| 4. Have you frequently banged into something, or felt any difficulty in writing characters, recently? | | | | The patient should be required to show spontaneous writing and be observed in the finger-to-nose test and heel-to-shin test and while walking (in a straight line by putting the heel of one foot in front of the toe of the other foot alternately). |

| Date: | month/ | date/ | year |
|---------|------------|----------|------|
| Subject | Identifica | ition Co | de: |

| Symptoms | Have you had significantly uexperience for following? | ınusual | If "yes," describe symptoms specifically | Objective test to be applied: results should be recorded in the Objective PML checklist |
|---|---|---|---|---|
| | Yes | No | | |
| 5. Have you often experienced an inability to understand wording someone has said recently? | | | | Ability to follow a series of instruction (stick out the tongue and touch the left ear with the left fingers while keeping the eyes closed). |
| 6. Do you have any continuous problems in your memory or thinking? | | | | The patient should be reminded of the 3 objects after 1 minute or longer distraction; ability to follow instructions |
| 7. Have you experienced continuous hypesthesia or other loss of sensation? | | | | Sensation should be tested<br>by neighboring needle<br>stimulation |

| Conducted by | y (signatuı | re or na | ame/sea | l) |
|--------------|-------------|----------|---------|----|
| sea1 | month/ | date/ | vear | |

Objective PML checklist

For a patient with subjective symptoms.

Please perform the tests for objective findings corresponding to the observed subjective symptoms.

| Date: | month/ | date/ | year |
|---------|------------|---------|------|
| Subject | Identifica | tion Co | de: |

| Positive subjective | Objective tests applied | Test 1 | esults | Brief description of the |
|---|---|---|---|---|
| symptoms | | Normal | Abnormal | observed abnormality |
| 1. Difficulty in vision and reading | Visual field and eye movement should be tested. | | | |
| 2. Difficulty in speech | Spontaneous observation should be performed for patient's speech for dysarthria or aphasia. The patient should be requested to answer names of some objects and to repeat some phrases with several words. | | | |
| 3. Muscle weakness in the upper or lower limb | Pronator deflection test (Barré procedure) and/or a test to see ability to keep the arm being rotated Ability to hop on one foot; to tap with the foot and finger. A symmetry test in the muscle. | | | |
| 4. Bang into something or difficulty in writing | The patient should be required to show spontaneous writing and observed in the finger-to-nose test and heel-to-shin test and while walking (in a straight line by putting the heel of one foot in front of the toe of the other foot alternately). | | | |

| Date: | month/ | date/ | year |
|---------|------------|----------|------|
| Subject | Identifica | ition Co | de: |

| Positive subjective symptoms | Objective tests applied | Test results | | Brief description of the |
|---|---|---|---|---|
| | | Normal | Abnormal | observed abnormality |
| 5. Difficulty in understanding others | Ability to follow a series of instruction (stick out the tongue and touch the left ear with the left fingers while keeping the eyes closed). | | | |
| 6. Problems in memory or thinking | The patient should be reminded of the 3 objects after 1 minute or longer distraction; ability to follow instructions | | | |
| 7.<br>Problems of hypesthesia | Sensation should be tested by neighboring needle stimulation | | | |

- The patient whose reported symptoms were confirmed in the Objective PML checklist should be instructed to visit a neurologist. The patient should be followed a week after the Objective PML checklist for confirmation of re-manifestation of the reported subjective symptoms.
- Any positive findings in the Objective PML checklist must be provided to the sponsor.

Conducted by (signature or name/seal)

seal month/date/ year

| Ap | pendix E – Follow-Up ( | Survey Form | | | |
|---|---|---|---|---|---|
| | | | Subject Identification Code: | | |
| | Number of months after the last dose of the study d | | | | |
| | | .□ 18 mo.□ 24 mo.□ | | | |
| | | | Date: | month/ | date/ year |
| 1. Have you been diagnosed with colon dysplasia (one of the precancerous lesions) or colon cancer, lymphoma, or other cancers since the last contact/visit in the study? | | | | | No<br>□ |
| If "y | ves," please answer to the follo | | · | | |
| • | Colon dysplasia | Yes/No | Date of the diagnosis: month/ date/ year | | |
| • | Colonic cancer | Yes/No | Date of the diagnosis: month/ date/ year | | |
| • | Lymphoma | Yes/No | Date of the diagnosis: month/ date/ year | | |
| • | Other: (Specify) | Yes/No | Date of the diagnosis: month/ date/ year | | |
| 2. Have you been diagnosed as having progressive multifocal leukoencephalopathy (also known as PML) since the last contact/visit in the study? | | | | | No |
| <u>If "y</u> | ves," please answer to the follo | wing question:. | | | |
| • | Date of the diagnosis: mon | th/ date/ year | | | |
| 3. Have you undergone an enterectomy since the last contact/visit in the study? | | | | Yes | No<br>□ |
| If "v | ves," please answer to the follo | wing questions:. | | | |
| • | Colectomy | Yes/No | Date of the diagnosis: month/ date/ year | | |
| • | Small bowel resection | Yes/No | Date of the diagnosis: month/ date/ year | | |
| | The following 3 question | ons will be comple | eted only once at 6 months after the last dose of the | study drug. | |
| 4. Have you been diagnosed as having an infection requiring hospitalization since the last study visit? | | | | | No |
| If "yes," please answer to the following questions:. | | | | | _ |
| Specify the reason for the hospitalization/diagnosis | | | | | |
| Reason: | | | | | |
| • | Date of the diagnosis: mon | th/ date/ year | | | |
| 5. For female patients: Have you become pregnant since the last study visit? | | | | | No<br>□ |
| <u>If "y</u> | ves," please answer to the follo | | | | |
| <ul> <li>The PREGNANCY REPORTING FORM should be completed</li> </ul> | | | | Not applicable | |
| • | Specify the estimated delive | ry date: month/ | date/ year | | |
| 6. | | • | me pregnant since the last study visit? | Yes | No<br>□ |
| If "y | ves," please answer to the follo | | | | |
| The PREGNANCY REPORTING FORM should be completed | | | | | plicable |
| Specify the estimated delivery date: month/ date/ year | | | | | Ш |
| | Investigator (signature or name/sea | | | | |
| | | | | | sea1 |
| | | | <u>mont</u> | h/ date | e/ year |